CLINICAL TRIAL: NCT04518410
Title: Adaptive Platform Treatment Trial for Outpatients With COVID-19 (Adapt Out COVID)
Brief Title: ACTIV-2: A Study for Outpatients With COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eli Lilly and Company (Industry); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); Brii Biosciences Limited (Industry); AstraZeneca (Industry); Sagent Pharmaceuticals (Industry); Synairgen Research Ltd. (Industry); Bristol-Myers Squibb (Industry); SAb Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5401/ACTIV-2; 38742 (Other: DAIDS-ES)
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Coronavirus; Covid19
Keywords: COVID-19; Coronavirus; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-2; ACTIV2
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Coronaviridae Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — bamlanivimab; cilgavimab and tixagevimab drug combination; camostat; ogalvibart, crexavibart drug combination; SAB-185; casirivimab and imdevimab drug combination; casirivimab; imdevimab; ogalvibart; crexavibart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Unblinded data will be provided to the Data and Safety Monitoring Board for interim analyses. Unblinded Day 28 data will also be provided to a small group of people from the company who owns the investigational agent, to assist the company in deciding if the agent should move into phase 3 evaluation; or in choosing a dose of their agent to move into phase 3 evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (25):
- Bamlanivimab 7000 mg (Phase 2) (Experimental): Administered by IV infusion.
  Interventions: Biological: bamlanivimab 7000mg
- Bamlanivimab 7000mg Placebo (Phase 2) (Placebo Comparator): Administered by IV infusion
  Interventions: Drug: Placebo for Bamlanivimab 7000mg
- Bamlanivimab 700mg (Phase 2) (Experimental): Administered by IV infusion
  Interventions: Biological: bamlanivimab 700mg
- Bamlanivimab 700mg Placebo (Phase 2) (Placebo Comparator): Administered by IV infusion
  Interventions: Drug: Placebo for Bamlanivimab 700mg
- Bamlanivimab 700mg (Phase 3) (Experimental): Administered by IV infusion
  Interventions: Biological: bamlanivimab 700mg
- BRII-196+BRII-198 (Pooled Phase 2/3) (Experimental): Administered by IV infusion
  Interventions: Biological: BRII-196+BRII-198
- BRII-196+BRII-198 Placebo (Pooled Phase 2/3) (Placebo Comparator): Administered by IV infusion
  Interventions: Drug: Placebo for BRII-196+BRII-198
- AZD7442 (IV) (Phase 2) (Experimental): Administered by IV infusion
  Interventions: Biological: AZD7442 (IV)
- AZD7442 (IV) Pooled Placebo (Phase 2) (Placebo Comparator): Administered by IV infusion; shared placebo includes AZD7442 (IM) placebo and placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for AZD7442 (IV)
- AZD7442 (IM) (Phase 2) (Experimental): Administered by IM injection
  Interventions: Biological: AZD7442 (IM)
- AZD7442 (IM) Pooled Placebo (Phase 2) (Placebo Comparator): Administered by IM injection; shared placebo includes AZD7442 (IV) placebo and placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for AZD7442 (IM)
- SNG001 (Phase 2) (Experimental): Administered by inhalation
  Interventions: Drug: SNG001
- SNG001 Pooled Placebo (Phase 2) (Placebo Comparator): Administered by inhalation; shared placebo includes placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for SNG001
- Camostat (Phase 2) (Experimental): Administered as oral tablets
  Interventions: Drug: Camostat
- Camostat Pooled Placebo (Phase 2) (Placebo Comparator): Administered as oral tablets; shared placebo includes placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for Camostat
- SAB-185 (low dose) (Phase 2) (Experimental): Administered by IV infusion
  Interventions: Biological: SAB-185 (3,840 Units/kg)
- SAB-185 (low dose) Pooled Placebo (Phase 2) (Placebo Comparator): Administered by IV infusion; includes SAB-185 (high dose) placebo and placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for SAB-185 (low dose)
- SAB-185 (low dose) (Phase 3) Non-OMICRON population (Experimental): Administered by IV infusion.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  Interventions: Biological: SAB-185 (3,840 Units/kg)
- Casirivimab and Imdevimab (Phase 3) Non-OMICRON population (Active Comparator): Administered by IV infusion.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  Interventions: Drug: CASIRIVIMAB + IMDEVIMAB
- SAB-185 (high dose) (Phase 2) (Experimental): Administered by IV infusion
  Interventions: Biological: SAB-185 (10,240 Units/kg)
- SAB-185 (high dose) Pooled Placebo (Phase 2) (Placebo Comparator): Administered by IV infusion; includes SAB-185 (low dose) placebo and placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for SAB-185 (high dose)
- BMS 986414+BMS 986413 (Phase 2) (Experimental): Administered as subcutaneous (SC) injections
  Interventions: Biological: BMS-986414 + BMS-986413
- BMS 986414+BMS 986413 Pooled Placebo (Phase 2) (Placebo Comparator): Administered as subcutaneous (SC) injections; shared placebo includes placebo from other comparator arms in the study.
  Interventions: Drug: Placebo for BMS-986414 + BMS-986413
- SAB-185 (low dose) (Phase 3) OMICRON population (Experimental): Administered by IV infusion The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  Interventions: Biological: SAB-185 (3,840 Units/kg)
- Casirivimab and Imdevimab (Phase 3) OMICRON population (Active Comparator): Administered by IV infusion The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  Interventions: Drug: CASIRIVIMAB + IMDEVIMAB

INTERVENTIONS:
Biological: bamlanivimab 7000mg — Administered by single IV infusion. Participants are no longer being randomized to this intervention.
  Other Names: LY3819253
  Arms: Bamlanivimab 7000 mg (Phase 2)
Biological: BRII-196+BRII-198 — 1000 mg (BRII-196)/1000 mg (BRII-198) combination therapy. Administered by consecutive IV infusions as single dose. Participants are no longer being randomized to this intervention.
  Arms: BRII-196+BRII-198 (Pooled Phase 2/3)
Biological: AZD7442 (IV) — 300 mg AZD7442 (150 mg AZD8895 + 150 mg AZD1061). Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  Other Names: AZD8895 + AZD1061
  Arms: AZD7442 (IV) (Phase 2)
Biological: AZD7442 (IM) — Administered intramuscularly as 2 separate injections sequentially (300 mg AZD8895 then 300 mg AZD1061) for one dose. Injections administered in the side of the thigh, one injection in each thigh. Participants are no longer being randomized to this intervention.
  Other Names: AZD8895 + AZD1061
  Arms: AZD7442 (IM) (Phase 2)
Drug: SNG001 — 1.3 mL solution administered once daily for 14 days using Aerogen Ultra nebulizer (inhalation device). Participants are no longer being randomized to this intervention.
  Arms: SNG001 (Phase 2)
Drug: Camostat — 200 mg (2 x 100 mg) film-coated tablets administered orally every 6 hours for 7 days. Participants are no longer being randomized to this intervention.
  Other Names: FOY-305; camostat mesilate; camostat mesylate
  Arms: Camostat (Phase 2)
Biological: BMS-986414 + BMS-986413 — Administered subcutaneously (SC) as 4 separate injections for one dose (two injections of C135-LS 200mg and two injections of C144-SL 200mg). Participants are no longer being randomized to this intervention.
  Other Names: C135-LS + C144-LS
  Arms: BMS 986414+BMS 986413 (Phase 2)
Biological: SAB-185 (3,840 Units/kg) — Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  Other Names: Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (Tc bovine-derived)
  Arms: SAB-185 (low dose) (Phase 2); SAB-185 (low dose) (Phase 3) Non-OMICRON population; SAB-185 (low dose) (Phase 3) OMICRON population
Biological: SAB-185 (10,240 Units/kg) — Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  Other Names: Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (Tc bovine-derived)
  Arms: SAB-185 (high dose) (Phase 2)
Drug: CASIRIVIMAB + IMDEVIMAB — 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
  Other Names: REGN10933 + REGN10987; REGN-COV2
  Arms: Casirivimab and Imdevimab (Phase 3) Non-OMICRON population; Casirivimab and Imdevimab (Phase 3) OMICRON population
Drug: Placebo for Bamlanivimab 7000mg — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: Bamlanivimab 7000mg Placebo (Phase 2)
Drug: Placebo for Bamlanivimab 700mg — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: Bamlanivimab 700mg Placebo (Phase 2)
Drug: Placebo for BRII-196+BRII-198 — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: BRII-196+BRII-198 Placebo (Pooled Phase 2/3)
Drug: Placebo for SNG001 — Trisodium citrate dihydrate, di-sodium hydrogen-phosphate, sodium dihydrogen-phosphate dihydrate, racemic methionine (DL-methionine) and water. 1.3 mL solution administered once daily for 14 days using Aerogen Ultra nebulizer (inhalation device). Participants are no longer being randomized to this intervention.
  Arms: SNG001 Pooled Placebo (Phase 2)
Drug: Placebo for Camostat — 200 mg (2 x 100 mg) film-coated tablets administered orally every 6 hours for 7 days. Participants are no longer being randomized to this intervention.
  Arms: Camostat Pooled Placebo (Phase 2)
Drug: Placebo for SAB-185 (low dose) — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: SAB-185 (low dose) Pooled Placebo (Phase 2)
Drug: Placebo for BMS-986414 + BMS-986413 — Administered SC as 4 separate injections for one dose. Participants are no longer being randomized to this intervention.
  Arms: BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Drug: Placebo for AZD7442 (IV) — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: AZD7442 (IV) Pooled Placebo (Phase 2)
Drug: Placebo for AZD7442 (IM) — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: AZD7442 (IM) Pooled Placebo (Phase 2)
Drug: Placebo for SAB-185 (high dose) — Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
  Arms: SAB-185 (high dose) Pooled Placebo (Phase 2)
Biological: bamlanivimab 700mg — Administered by single IV infusion. Participants are no longer being randomized to this intervention.
  Other Names: LY3819253
  Arms: Bamlanivimab 700mg (Phase 2); Bamlanivimab 700mg (Phase 3)

SUMMARY:
Drug studies often look at the effect one or two drugs have on a medical condition, and involve one company. There is currently an urgent need for one study to efficiently test multiple drugs from more than one company, in people who have tested positive for COVID-19 but who do not currently need hospitalization. This could help prevent disease progression to more serious symptoms and complications, and spread of COVID-19 in the community.

This study looks at the safety and effectiveness of different drugs in treating COVID-19 in outpatients. In Phase II, participants in the study will be treated with either a study drug or with placebo. In protocol version 7.0, participants in Phase III of the study will be treated with either a study drug or active comparator drug. Participants assigned to the bamlanivimab agent/placebo arm and will have 28 days of intensive follow-up following study drug administration, followed by limited follow-up through 24 weeks in phase II and in phase III. All other investigational agents and their corresponding placebo arms will involve 28 days of intensive follow-up, followed by limited follow-up through 72 weeks in phase II and phase III. Additional study visits may be required, depending on the agent.

DETAILED DESCRIPTION:
This is a master protocol to evaluate the safety and efficacy of multiple investigational agents aimed at modifying the host immune response to SARS-CoV-2 infection, or directly enhancing viral control in order to limit disease progression.

The study includes both infused and non-infused agents and is a randomized controlled platform that allows agents to be added and dropped during the course of the study for efficient phase II and phase III testing of new agents within the same trial infrastructure.

Version 7 of the protocol provided for blinded phase II evaluation of an investigational agent for superiority to placebo among participants at lower risk of progression to hospitalization or death, regardless of the mode of administration of the agent.

Agents that graduate to phase III after initiation of the protocol version will be evaluated in persons at higher risk for progression to hospitalization or death for non-inferiority to an active comparator (monoclonal antibody cocktail of casirivimab plus imdevimab (REGEN-COV, Regeneron). This active comparator has been shown to be effective in this population in preventing hospitalization or death. When two or more agents are being evaluated in the same phase of the study, the trial design includes sharing of the control group (placebo in phase II and active comparator in phase III) for efficient evaluation of each agent.

Investigational agents will be approved by the Trial Oversight Committee (TOC) for phase II evaluation based on the presence of in vitro data demonstrating promise as anti-SARS-CoV-2 therapeutics in pre-clinical testing, and for which there are suitable pharmacokinetics and safety data from phase I testing, or through clinical or research testing for a different indication, and agent availability. Investigational agents will be included in phase III evaluation based on agent entry criteria for phase III as outlined in the protocol (or by TOC approval based on data available outside ACTIV-2).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Documentation of laboratory-confirmed SARS-CoV-2 infection, as determined by a molecular (nucleic acid) or antigen test from any respiratory tract specimen (e.g. oropharyngeal, nasopharyngeal (NP), or nasal swab, or saliva) collected ≤240 hours (10 days) prior to study entry. Laboratory-confirmed SARS-CoV-2 infection outside the US must be conducted at a DAIDS-approved laboratory.
* Able to begin study treatment no later than 7 days from self-reported onset of COVID-19 related symptom(s) or measured fever, where the first day of symptoms is considered symptom day 0 and defined by the self-reported date of first reported sign/symptom from the following list:

  * subjective fever or feeling feverish
  * cough
  * shortness of breath or difficulty breathing at rest or with activity
  * sore throat
  * body pain or muscle pain/aches
  * fatigue
  * headache
  * chills
  * nasal obstruction or congestion
  * nasal discharge
  * loss of taste or smell
  * nausea or vomiting
  * diarrhea
  * temperature > 38°C (100.4°F)
* One or more of the following signs/symptoms within 24 hours of participating in the study:

  * subjective fever or feeling feverish
  * cough
  * shortness of breath or difficulty breathing at rest or with activity
  * sore throat
  * body pain or muscle pain/aches
  * fatigue
  * headache
  * chills
  * nasal obstruction or congestion
  * nasal discharge
  * loss of taste or smell
  * nausea or vomiting
  * diarrhea
  * temperature > 38°C (100.4°F)
* Oxygen levels of ≥92% obtained at rest (adjusted as needed for altitude) by study staff within 24 hours of study entry. For a potential participant who regularly receives chronic supplementary oxygen for an underlying lung condition, their oxygen saturation should be measured while on their standard home oxygen supplementation level.
* Participant must agree not to participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period until hospitalization or 28 days after the start of the study, whichever occurs first.
* Meet the protocol definition of being at "higher" risk of progression to hospitalization or death (BRII-196/BRII-198).
* In Phase III, meeting the protocol definition of being at "higher" risk of progression to hospitalization or death (SNG001, SAB-185, BMS 986414+BMS 986413)
* For participants of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to study entry by any clinic or laboratory that has a CLIA certification or its equivalent, or by a point of care (POC)/CLIA-waived test. Note: Participants not of reproductive potential are eligible without requiring the use of a contraceptive method (BRII-196/BRII-198. AZD7442 [IV], AZD7442 [IM], SNG001, Camostat, SAB-185, BMS 986414+BMS 986413).
* Participants that engage in sexual activity that may lead to pregnancy in their partner must agree to either remain abstinent or use male contraceptives. They are strongly advised to inform their non-pregnant sexual partners of reproductive potential to use effective contraceptives for 24 weeks after investigational product is administered. Participants with pregnant partners should use condoms during vaginal intercourse through 24 weeks after investigational agent administration. Participants should refrain from sperm donation for 24 weeks after investigational agent administration (BRII-196/BRII-198, AZD7442 [IV], AZD7442 [IM], SAB-185).
* Participants that engage in sexual activity that may lead to pregnancy in their partner must agree to either remain abstinent or use male contraceptives for 30 days after investigational agent administration. They are also strongly advised to inform their non-pregnant sexual partners of reproductive potential to sue effective contraceptives for 30 days after investigational agent is administered to the participant. Participants with pregnant partners should use condoms during vaginal intercourse through 30 days after last dose of investigational agent administration. Participants should refrain from sperm donation for 30 days after investigational agent administration (SNG001).
* Participants that engage in sexual activity that may lead to pregnancy in their partner must agree to either remain abstinent or use male contraceptives. They are also strongly advised to inform their non-regnant sexual partners of reproductive potential to use effective contraceptives from study entry through 90 days after study treatment. Participants with pregnant partners should use condoms during vaginal intercourse from study entry through 90 days after the last dose of the study treatment. Participants should refrain from sperm donation from study entry through 90 days after the last dose of study treatment (Camostat).
* If participating in sexual activity that could lead to pregnancy, participants who are of reproductive potential must agree to use effective contraception for 24 weeks after investigational agent is administered. This would include oral contraceptives, implanted contraceptives, implanted contraceptives, intrauterine devices, and barrier methods.
* If participating in sexual activity that could lead to pregnancy, participants who are of reproductive potential must agree to use highly effective contraception for 24 weeks after investigational agent is administered (AZD7442 [IV], AZD7442 [IM], SAB-185).
* If participating in sexual activity that could lead to pregnancy, participants who are of reproductive potential must agree to use effective contraception for 30 days after investigational agent is administered (SNG001).
* If participating in sexual activity that could lead to pregnancy, participants who are of reproductive potential must agree to use effective contraception for 90 days after the last dose of treatment (Camostat).
* If participating in sexual activity that could lead to pregnancy, participants who are of reproductive potential must agree to use highly effective contraception for at least 48 weeks after the investigational agent is administered (BMS 986414+BMS 986413).

Exclusion Criteria:

* History of or current hospitalization for COVID-19.
* For the current SARS-CoV-2 infection, any positive SARS-CoV-2 nucleic acid or antigen tests from any respiratory tract specimen collected > 240 hours prior to study entry.
* Current need for hospitalization or immediate medical attention.
* Use of any prohibited medication listed in the protocol and/or use of systemic or inhaled steroids for the purpose of COVID-19 treatment (new or increased dose from chronic baseline) within 30 days prior to study.
* Receipt of convalescent COVID-19 plasma or other antibody-based anti-SARS-CoV-2 treatment or prophylaxis at any time prior to study entry.
* Receipt of other investigational treatments for SARS-CoV-2 any time before participating in the study (not including drugs approved and taken for other conditions/diseases or COVID-19 vaccines).
* Known allergy/sensitivity or hypersensitivity to study drug or placebo.
* Any condition requiring surgery up to 7 days before participating in the study, or that is considered life threatening up to 30 days before participating in the study.
* Currently pregnant or breastfeeding (BRII-196/BRII-198, AZD7442 [IV], AZD7442 [IM], SNG001, Camostat, SAB-185, BMS 986414+BMS 986413).
* In phase II, meeting the protocol definition of being at "higher" risk of progression to hospitalization or death (AZD7442 [IV], AZD7442 [IM], SNG001, Camostat, SAB-185, BMS 986414+BMS 986413).
* Inflammatory skin conditions that compromise the safety of intramuscular (IM) injections, or other overlying skin conditions or tattoos that would preclude the assessment of injection site reactions, per the discretion of the investigator (AZD7442 [IM]).
* Inflammatory skin conditions that compromise the safety of subcutaneous (SC) injections, or other overlying skin conditions or tattoos that would preclude the assessment of infection site reactions, per the discretion of the investigator (BMS 986414+BMS 986413).
* History of coagulopathy which, in the opinion of the investigator, would preclude IM injection, or use of oral or injectable anticoagulants (protocol provides more information on prohibited medications) (AZD7442 [IM]).
* Use of or need for chronic supplemental oxygen (SNG001).
* Known severe liver disease prior to enrollment (defined as ALT or AST > 5 times upper limit of normal or end stage liver disease with Child-Pugh Class C or Child-Pugh-Turcotte score ≥ 10) (Camostat).
* Known severe kidney disease prior to enrollment (defined as estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m² or on renal-replacement therapy such as peritoneal dialysis or hemodialysis (Camostat)

Other investigational drug protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4044 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, MAS, Study Chair — University of California, San Diego
Locations (252):
- United States (207):
  - Pinnacle Research Group (Site 1082), 321 E. 10th Street, Anniston, Alabama
  - North Alabama Research Center LLC (Site 1194), 721 W. Market St., Ste. B, Athens, Alabama
  - University of Alabama at Birmingham (Site 1005), 908 20th Street South, Birmingham, Alabama
  - Cullman Clinical Trials (Site 1140), 501 Clark St. NE., Cullman, Alabama
  - Jasper Summit Research, LLC. (Site 1056), 1280 Summit, Jasper, Alabama
  - Absolute Clinical Research, LLC. (Site 1186), 7725 North 43rd Avenue, Ste. 211, Phoenix, Arizona
  - University of Arizona (Site 1043), 1501 N. Campbell Ave., Rm. 6410, Tucson, Arizona
  - Omnibus Clinical Research (Site 1253), 3340 W. Ball Road, Ste. I, Anaheim, California
  - Franco A. Felizarta MD (Site 1174), 3535 San Dimas St., Bakersfield, California
  - Clearview Medical Research LLC. (Site 1251), 2714 Hidaway Ave., Ste. 103, Canyon Country, California
  - St. Jude Heritage Medical Group (Site 1093), 2151 N. Harbor Blvd., Fullerton, California
  - University of California San Diego (Site 1160), 9350 Campus Point Drive, Perlman Cancer Cancer, La Jolla, California
  - Fadi A. Haddad, MD, Inc. (Site 1146), 8860 Center Dr., Ste. 320, La Mesa, California
  - Atella Clinical Research (Site 1111), 5451 La Palma Avenue, La Palma, California
  - Loma Linda University Health (Site 1110), 11374 Mountain View, Dover Bldg, Ste. C, Loma Linda, California
  - University of Southern California (Site 1057), 1300 N. Mission Rd., Rm 349, Los Angeles, California
  - UCLA CARE Center (Site 1003), 11075 Santa Monica Blvd., Suite 100, Los Angeles, California
  - Science 37, Inc. (Site 1124), 12121 Bluff Creek Dr., Ste. 100, Los Angeles, California
  - VA Northern California Health Care System (NAVREF) (Site 1137), 10535 Hospital Way, Mather, California
  - Central Valley Research, LLC (Site 1085), 400 E. Orangeburg Ave., Ste. 5, Modesto, California
  - Hoag Memorial Hospital Presbyterian (Site 1200), 1 Hoag Dr., Newport Beach, California
  - Valley Clinical Research, Inc. (Site 1059), 18433 Roscoe Blvd., Ste 210, Northridge, California
  - University of California Irvine (Site 1083), 843 Health Sciences Road, Orange, California
  - FOMAT Medical Research (Site 1136), 300 South A Street, Oxnard, California
  - Eisenhower Medical Center (Site 1040), 39000 Bob Hope Drive, Rancho Mirage, California
  - Paradigm Research (Site 1150), 3652 Eureka Way, Redding, California
  - Riverside Medical Clinic (Site 1232), 7117 Brockton Ave., Riverside, California
  - University of California Davis Medical Center (Site 1097), 2315 Stockton Blvd., Sacramento, California
  - Premier Urgent Care Centers of California, Inc. (Site 1176), 284 E. Highland Ave., San Bernardino, California
  - University of California San Diego (Site 1002), 220 Dickinson Street, San Diego, California
  - Zion Medical Center (Site 1063), 4647 Zion Avenue, San Diego, California
  - VA San Diego Health System (Stie 1127), 3350 La Jolla, San Diego, California
  - University of California San Francisco (Site 1009), 995 Potrero Ave., Building 80, Ward 84, San Francisco, California
  - San Francisco Research Institute (Site 1210), 2435 Ocean Ave., San Francisco, California
  - Stanford University (Site 1213), 1201 Welch Road, Stanford, California
  - Millennium Clinical Trials (Site 1260), 550 Saint Charles Dr., Ste. 208, Thousand Oaks, California
  - Office of Ramesh V. Nathan, MD (Site 1073), 2220 Lynn Rd., Ste. 301, Thousand Oaks, California
  - Harbor UCLA (Site 1022), 1124 West Carson Street, Torrance, California
  - Allianz Research Institute Inc. (Site 1159), 14120 Beach Blvd., Ste. 101, Westminster, California
  - University of Colorado (Site 1007), 12401 East 17th Avenue, Aurora, Colorado
  - UConn - Institute for Collaboration on Health (Site 1169), 2006 Hillside Rd., Unit 1248, Storrs, Connecticut
  - Whitman-Walker Health (Site 1027), 1337 R Street NW., Washington D.C., District of Columbia
  - Imagine Research of Palm Beach County (Site 1157), 709 S. Federal Hwy., Ste. 2, Boynton Beach, Florida
  - Bradenton Research Center Inc. (Site 1109), 3924 9th Ave. W, Bradenton, Florida
  - Synergy Healthcare (Site 1099), 300 Riverside Drive E., Ste. 1350, Bradenton, Florida
  - Cardiology Physicians, P.A. (Site 1180), 305 Memorial Medical Pkwy., Ste. 301, Daytona Beach, Florida
  - Midland Florida Clinical Research Center LLC (Site 1130), 665 Peachwood Drive, DeLand, Florida
  - Integrity Clinical Research (Site 1214), 3901 NW 79th Ave., Doral, Florida
  - Universal Axon Clinical Research (Site 1077), 3650 NW 82nd Ave., Doral, Florida
  - EMINAT Research (Site 1202), 2500 E. Commercial Blvd., Fort Lauderdale, Florida
  - Holy Cross Health (Site 1072), 4725 North Federal Highway, Fort Lauderdale, Florida
  - North Florida / South Georgia Veterans Health System (Site 1133), 1601 SW Archer Rd., Gainesville, Florida
  - University of Florida (Site 1047), 1600 SW. Archer Rd., Gainesville, Florida
  - NW FL Clinical Research Group, LLC. (Site 1046), 400 Gulf Breeze Parkway, Gulf Breeze, Florida
  - Indago Research and Health Center (Site 1050), 3700 W. 12th Ave., Ste. 300, Hialeah, Florida
  - AGA Clinical Trials (Site 1026), 900 West 49th Street, Hialeah, Florida
  - Community Research of South Florida (Site 1197), 7100 W. 20th Ave., Ste. 403, Hialeah, Florida
  - New Generation Medical Research (Site 1204), 7600 W. 20th Ave., Ste. 106, Hialeah, Florida
  - Best Quality Research, Inc. (Site 1237), 2387 W. 68th St., Ste. 403, Hialeah, Florida
  - Innovative Health Medical Center (Site 1222), 6750 Taft Street, Hollywood, Florida
  - University of Florida Jacksonville (Site 1039), 655 West 8th Street, Jacksonville, Florida
  - Mayo Clinic Jacksonville (Site 1149), 4500 San Pablo Rd. S., Jacksonville, Florida
  - Gonzalez MD & Aswad MD Health Services (Site 1238), 3401 NW. 7th Street, Miami, Florida
  - Clintex Research Group, Inc. (Site 1231), 590 SW. 27th Ave., Miami, Florida
  - Advance Medical Research Center (Site 1193) 330 SW. 27th Ave., Ste. 701, Miami, Florida
  - University of Miami Miller School of Medicine CoVID Unit (Site 1068), 1425 NW. 10th Ave., Miami, Florida
  - Florida International Medical Research (Site 1239), 1890 S. Red Rd., Ste. 103, Miami, Florida
  - D&H National Research Centers (Site 1205), 8485 Bird Road, Miami, Florida
  - Allied Biomedical Research Institute (Site 1227), 7100 SW. 47th St., Ste. 220, Miami, Florida
  - Miami Clinical Research (Site 1089), 2400 SW. 69th Ave., Miami, Florida
  - Research Institute of South Florida, Inc. (Site 1201), 9835 SW. 72nd Street, Ste. 201, Miami, Florida
  - RM Medical Research, Inc. (Site 1230), 10346 W. Flagler St., Miami, Florida
  - Pro Live Medical Research Corp (Site 1219), 12781 SW. 42nd Street, Miami, Florida
  - Miami Dade Medical Research Institute, LLC (Site 1223), 8955 SW. 87th Ct., Miami, Florida
  - QC Trials (Site 1117), 300 W. 41st Street, Ste. 203, Miami Beach, Florida
  - Lakes Research (Site 1037), 5801 NW 151 Street, Miami Lakes, Florida
  - Savin Medical Group, LLC. (Site 1212), 5789B NW. 151st Street, Miami Lakes, Florida
  - Amber Clinical Research, LLC. (Site 1206), 9000 NE. 2nd Avenue, Miami Shores, Florida
  - Bravo Health Care Center (Site 1221), 1440 79 Street, North Bay Village, Florida
  - Orlando Immunology Center (Site 1045), 1707 North Mills Avenue, Orlando, Florida
  - Clintheory (Site 1203), 7350 Sandlake Commons Blvd., Orlando, Florida
  - IMIC, Inc. (Site 1141), 18320 Franjo Rd, Palmetto Bay, Florida
  - Family Clinical Trials (Site 1236), 1601 N. Palm Ave., Ste. 102, Pembroke Pines, Florida
  - Physician Care Clinical Research, LLC. (Site 1242), 1617 S. Tuttle Ave., Ste. 1A, Sarasota, Florida
  - Bassetti Medical Research, Inc. (Site 1158), 5825 US Highway 27 N., Sebring, Florida
  - DBC Research (Site 1188), 7707 N. University Dr., Ste. 106, Tamarac, Florida
  - ETNA Medical Center (Site 1225), 7401 N. University Drive, Tamarac, Florida
  - Moore Clinical Research, Inc. (Site 1164), 4257 W. Kennedy Blvd., Tampa, Florida
  - Tampa General Hospital Family Care Center Healthpark (Site 1088), 5802 N. 30th Street, Tampa, Florida
  - Infectious Disease Consultants of the Treasure Coast (Site 1171), 3735 11th Cir., Ste. 201, Vero Beach, Florida
  - AIDS Research and Treatment Center of the Treasure Coast (Site 1095), 981 37th Place, Vero Beach, Florida
  - Triple O Research Institute PA (Site 1121), 2580 Metrocentre Blvd., Ste. 4, West Palm Beach, Florida
  - The Ponce de Leon Center (site 1015), 341 Ponce De Leon Avenue Northeast, Atlanta, Georgia
  - Rare Disease Research, LLC. (Site 1248), 1891 Howell Mill Rd.NW, Ste. B, Atlanta, Georgia
  - Agile Clinical Rsearch Trials, LLC (Site 1051), 750 Hammond Drive, Atlanta, Georgia
  - Balanced Life Health Care Solutions/SKYCRNG (Site 1191), 2033 Buford Hwy., Ste. 109, Buford, Georgia
  - IACT Health (Site 1035), 800 Talbotton Road, Columbus, Georgia
  - Clintheory (Site 1254), 4300 Pleasant Hill Road, Duluth, Georgia
  - One Health Research Clinic, Inc. (Site 1250), 5880 Live Oak Pkwy, Ste. 160, Norcross, Georgia
  - Renew Health Clinical Research, LLC. (Site 1161), 1550 Janmar Rd., Snellville, Georgia
  - John A. Burns School of Medicine UH Clinics at Kakaako (Site 1177), 651 Ilalo St., Honolulu, Hawaii
  - Snake River Research, PLLC (Site 1120), 2900 Cortez Ave., Idaho Falls, Idaho
  - Metro Infectious Disease Consultants (Site 1106), 901 McClintock Dr., Ste. 201, Burr Ridge, Illinois
  - Chicago Clinical Research Institute (Site 1132), 611 W. Roosevelt Rd., Chicago, Illinois
  - Northwestern University (Site 1025), 645 North Michigan Ave, Chicago, Illinois
  - Rush University Medical Center (Site 1017), 600 Paulina St., Chicago, Illinois
  - University of Illinois at Chicago (Site 1147), 835 South Wood Street, Chicago, Illinois
  - University of Chicago (Site 1064), 5841 S. Maryland Ave., Chicago, Illinois
  - Great Lakes Clinical Trials (Site 1049), 5149 N. Ashland Ave., Chicago, Illinois
  - Investigators Research Group, LLC. (Site 1170), 321 E. Northfield Dr., Ste. 100, Brownsburg, Indiana
  - Roudebush VA Medical Center (Site 1217), 550 University Blvd, Indianapolis, Indiana
  - University of Kansas Medical Center (Site 1042), 3901 Rainbow Boulevard, Kansas City, Kansas
  - MedPharmics (Site 1065), 3800 Houma Blvd., Metairie, Louisiana
  - Clinical Trials of America, LLC. (Site 1245) 3201 Armand Street, Monroe, Louisiana
  - New Orleans Adolescent Trials Unit (Site 1028), 1440 Canal St., Suite 904, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center (Site 1153), 2000 Canal Street, New Orleans, Louisiana
  - Ochsner Clinic Foundation (Site 1218), 1514 Jefferson Highway, New Orleans, Louisiana
  - Baltimore VA Medical Center (Site 1258), 10 N. Greene St., Baltimore, Maryland
  - Johns Hopkins University (Site 1006), 1830 East Monument Street, Baltimore, Maryland
  - Walter Reed Army Institute of Research (Site 1118), 503 Robert Grant Ave., Silver Spring, Maryland
  - Massachusetts General Hospital (Site 1016), 55 Fruit Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 1166), 110 Francis Street, Boston, Massachusetts
  - Brigham and Women's Hospital - Therapeutics Clinical Research Site (Site 1023), 75 Francis Street, Boston, Massachusetts
  - University of Massachusetts Medical School (Site 1054), 55 Lake Avenue N., Worcester, Massachusetts
  - Vida Clinical Studies (Site 1244), 3815 Pelham Street, Dearborn, Michigan
  - Revive Research Institute (Site 1257), 32255 Northwestern Hwy., Farmington Hills, Michigan
  - Revival Research Corporation (Site 1256), 13409 East 14 Mile Road, Sterling Heights, Michigan
  - Memorial Hospital at Gulfport (Site 1104), 4500 13th Street, Gulfport, Mississippi
  - MedPharmics, LLC. (Site 1032), 15190 Community Rd., Gulfport, Mississippi
  - University of Missouri Health Care System (Site 1224), 1 Hospital Drive, Columbia, Missouri
  - Hannibal Clinic (Site 1129), 100 Medical Drive, Hannibal, Missouri
  - Washington University School of Medicine (Site 1008), 620 South Taylor, Suite 200, St Louis, Missouri
  - Bozeman Health Deaconess Hospital (Site 1115), 931 Highland Blvd, Ste. 3103, Bozeman, Montana
  - Mercury Street Medical Group (Site 1074), 300 W. Mercury St., Butte, Montana
  - Quality Clinical Research (Site 1112), 10040 Regency Circle, Omaha, Nebraska
  - Las Vegas Medical Research (Site 1048), 8530 W. Sunset Rd., Las Vegas, Nevada
  - AXCES Research Group (Site 1152), 531 Harkle Road, Santa Fe, New Mexico
  - Maimonides Medical Center (Site 1138), 4802 10th Avenue, Brooklyn, New York
  - University at Buffalo, Emergency Medicine (Site 1172), 77 Goodell Street, Buffalo, New York
  - Flushing Hospital Medical Center (Site 1067), 4500 Parsons Blvd, Flushing, New York
  - Jamaica Hospital Medical Center (Site 1066), 8900 Van Wyck Expressway, Jamaica, New York
  - Columbia Partnership for Prevention and Control of HIV/AIDS CTU (Site 1019), Columbia University Irving Medical Center, Department of Medicine - Division of Infectious Diseases, 180 Fort Washington Avenue, HP6 - Rm 604, New York, New York
  - Cornell Clinical Trials Unit (Site 1011), NewYork-Presbyterian Hospital-Weill Cornell Medical Center, 525 East 68th Street, New York, New York
  - Canton-Potsdam Hospital (Site 1076), 50 Leroy Street, Potsdam, New York
  - University of Rochester (Site 1010), 601 Elmwood Ave, Rochester, New York
  - SUNY Stony Brook NICHD (Site 1094), HSC L-02, Rm. 142 C, Stony Brook, New York
  - Bronx Prevention Research Center (Site 1108), 390 East 158th Street, The Bronx, New York
  - Lincoln Hospital (Site 1092), 249 East 149th Street, The Bronx, New York
  - Urban Health Plan, Inc. (Site 1243), 1065 Southern Blvd, The Bronx, New York
  - Jacobi Medical Center (Site 1105), 1400 Pelham Parkway South, The Bronx, New York
  - James J. Peters VA Medical Center (Site 1053), 130 West Kingsbridge Road, The Bronx, New York
  - University of North Carolina at Chapel Hill (Site 1001), 130 Mason Farm Rd., Bioinformatics Bldg, 2nd Floor, Chapel Hill, North Carolina
  - Carolina Clinical Research (Site 1167), 9040 Nations Ford Rd., Charlotte, North Carolina
  - Research Carolina Elite (Site 1247), 7480 Waterside Loop Road, Suite 201, Denver, North Carolina
  - Duke University Medical Center (Site 1041), 40 Duke Medicine Circle, Durham, North Carolina
  - Carteret Medical Group, LLC. (Site 1249), 302 Medical Park Ct., Morehead City, North Carolina
  - Wake Forest University Health Sciences (Site 1038), 1 Medical Center Boulevard, Winston-Salem, North Carolina
  - Sanford Health (Site 1084), 801 Broadway N., Fargo, North Dakota
  - The Christ Hospital (Site 1119), 2123 Auburn Avenue, Cincinnati, Ohio
  - Case Western Reserve University (Site 1033), 2061 Cornell Road, Cleveland, Ohio
  - MetroHealth Medical Center (Site 1195), 2500 Metrohealth Dr., Cleveland, Ohio
  - Ohio State University Medical Center (Site 1020), 480 Medical Center Drive, Columbus, Ohio
  - Cincinnati CRS (Site 1004), University of Cincinnati, University Hospital, 200 Albert Sabin Way, Ohio City, Ohio
  - STAT Research (Site 1107), 66 Remick Blvd., Springboro, Ohio
  - Ascension St. John Clinical Research Institute (Site 1090), 1725 East 19th Street, Tulsa, Oklahoma
  - Providence Portland Medical Center (Site 1098), 4805 NE. Glisan Street, Portland, Oregon
  - Kaiser Permanente Center for Health Research (Site 1079), 3800 N. Interstate Ave., Portland, Oregon
  - Portland VA Medical Center (Site 1131), 3710 SW US Veterans Hospital Rd., Portland, Oregon
  - Oregon Health and Science University (Site 1259), 3181 SW. 10th Avenue, Portland, Oregon
  - Doylestown Hospital (Site 1122), 595 W. State Street, Doylestown, Pennsylvania
  - University of Pennsylvania (Site 1031), 3400 Spruce Street, Philadelphia, Pennsylvania
  - The University of Pittsburgh (Site 1018), 3471 5th Ave., Pittsburgh, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System (Site 1070), University Drive C., Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (1142), 164 Summit Avenue, Providence, Rhode Island
  - Medtrial, LLC (Site 1134), 1718 Saint Julian Pl., Ste. 2, Columbia, South Carolina
  - Clinovacare Medical Clinical Research Center (Site 1211), 160 Medical Circle Suite D, West Columbia, South Carolina
  - American Indian Clinical Trials Research Network (Site 1148), 717 Meade Street, Rapid City, South Dakota
  - Sanford USD Medical Center (Site 1078), 1305 W. 18th St., Sioux Falls, South Dakota
  - Clinical Trials Center of Middle Tennessee (Site 1183), 100 Covey Drive, Franklin, Tennessee
  - Vanderbilt Therapeutics Clinical Research (Site 1013), Vanderbilt Health One Hundred Oaks, 719 Thompson Ln., Ste 47183, Nashville, Tennessee
  - Saint Hope Foundation Inc. (Site 1100), 6800 West Loop Street, Ste. 560, Bellaire, Texas
  - South Texas Medical Research Institute, Inc./TTS Research (Site 1198), 1420 River Road, Boerne, Texas
  - PanAmerican Clinical Research, LLC. (Site 1069), 1416 Palm Blvd., Brownsville, Texas
  - Trinity Health and Wellness Center (Site 1030), 219 Sunset Avenue, Dallas, Texas
  - UT Southwestern HIV/ID Clinical Trials Unit (Site 1208), 1936 Amelia Court, Dallas, Texas
  - Doctors Hospital at Renaissance Health Institute for Research and Development (Site 1145), 5323 S. McColl Rd., Edinburg, Texas
  - Sealy Institute for Vaccine Sciences Clincial Trials Program (Site 1044), 400 Harborside Drive, Galveston, Texas
  - Rheumatology Center of Houston (Site 1252), 1200 Binz St., Ste. 1495, Houston, Texas
  - Lyndon B. Johnson Hospital (Site 1014), 5656 Kelley Street, Houston, Texas
  - University of Texas Health Science Center at Houston (Site 1055), 6431 Fannin Street, Ste. 2.112, Houston, Texas
  - Houston Methodist Hospital (Site 1123), 6565 Fannin Street, Houston, Texas
  - Dynamic Medical Research Group (Site 1081), 8314 Southwest Fwy, Houston, Texas
  - Fairway Medical Clinic (Site 1156), 4910 Telephone Road, Houston, Texas
  - Houston Heart and Vascular Associates (Site 1215), 1485 FM 1960 Bypass R. E., Ste. 100, Humble, Texas
  - SMS Clincial Research, LLC. (Site 1060), 1210 N. Galloway Ave., Mesquite, Texas
  - Epic Medical Research, LLC (Site 1233), 106 Plaza Drive, Red Oak, Texas
  - San Antonio Military Medical Center (Site 1173), 3551 Roger Brooke Dr., San Antonio, Texas
  - Inova Fairfax Medical Campus (Site 1029), 3300 Gallows Road, Falls Church, Virginia
  - Clinical Research Partners LLC (Site 1196), 7110 Forest Ave., Ste. 201, Richmond, Virginia
  - EvergreenHealth (Site 1080), 12040 NE 128th Street, Ste MS-77, Kirkland, Washington
  - University of Washington ACTU (Site 1012), Harborview Medical Center, 325 9th Ave., Seattle, Washington
  - Providence Medical Research Center (Site 1075), 105 W. 8th Ave., Ste. 6050W, Spokane, Washington
  - Hershel Woody Williams VA Medical Center (Site 1128), 1540 Spring Valley Drive, Huntington, West Virginia
  - West VA University, Mary Babb Randolph Cancer Center (Site 1178), 1 Medical Center Drive, Morgantown, West Virginia
  - Vida Clinical Studies (Site 1246), 5757 West Oklahoma Avenue, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Inc. (Site 1036), 8701 Watertown Plank Road, Milwaukee, Wisconsin
  - Allegiance Research Specialists (Site 1162), 2645 N. Mayfair Rd., Ste. 200, Wauwatosa, Wisconsin
- Argentina (7):
  - Instituto Médico Platense (Site 3011), Avenida 51 335, La Plata, Buenos Aires
  - Fundación Sanatorio Güemes (Site 3001), Francisco Acuña de Figueroa 1240, Buenos Aires, Buenos Aires F.D.
  - Instituto Médico Río Cuarto (Site 3005), Hipólito Yrigoyen 1020, Río Cuarto, Córdoba Province
  - Instituto Médico de la Fundación Estudios Clínicos (Site 3009), Italia 428, Rosario, Santa Fe Province
  - Clínica Adventista Belgrano (Site 3007), Estomba 1710, Buenos Aires
  - Instituto Ave Pulmo (Site 3006), Carlos M. Alvear 3345, Mar del Plata
  - Hospital Universitario Austral (Site 3004), Av. Juan Domingo Peron, Derqui, Pilar
- Brazil (8):
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda (Site 4008), SGAS 613, Conjunto E, Lote 95, Sala 6, Brasília, Federal District
  - Hospital Das Clinicas Da Universidade Federal de Minas Gerais (Site 4001), Avenida Alfredo Balena 190, Belo Horizonte, Minas Gerais
  - SOM Federal University Minas Gerais Brazil (Site 4002), Avenida Alfredo Balena 190, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora da Conceicao (Site 4004), Avenida Francisco Trein 596, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão (Site 4007), Rua Engenheiro Paul Werner, 1141, Blumenau, Santa Catarina
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto (Site 4003), Avenida Bandeirantes 3900, Campus Universitário, Ribeirão Preto, São Paulo
  - Instituto de Pesquisa Clínica Evandro Chagas (Site 4005), Avenida Brasil, 4365, Rio de Janeiro
  - Hospital E Maternidade Celso Pierro (Site 4006), Avenue John Boyd Dunlop S/n, São Paulo
- Medical Arts Health Research Group (Site 2003), 360-1855 Kirschner Rd., Kelowna, British Columbia, Canada
- Centro Medico Militar (Site 9401), Finca El Palomar, Acatan, Sta. Rosita Zona 16, Guatemala City, Guatemala
- Mexico (8):
  - CIMAB SA de CV (Site 6002), Francisco I Madero 270 Sur, Torreón, Coahuila
  - Instituto Jalisciense de Investigacion Clinica SA de CV (Site 6005), Penitenciaria Numero 20, Colonia Centro, Guadalajara, Jalisco
  - Centro de Investigación Farmacéutica Especializada de Occidente (Site 6006), Av. Vallarta 1670, Piso 2 PH1, Colonia Americana, Guadalajara, Jalisco
  - Oaxaca Site Management Organization (Site 6004), Calle Humboldt 302, Colonia Centro, Oaxaca, Mexico City
  - Neurociencias Estudios Clinicos S.C. (Site 6008), Boulevard Alfonso G. Calderon, 2193 int 2 A desarrollo urbano 3 rios, Culiacán, Sinaloa
  - Hospital Civil De Culiacan (Site 6011), Avenida Álvaro Obregón 1422, Culiacán, Sinaloa
  - Eme Red Hospitalaria (Site 6010), Calle 33 No. 496, Mérida, Yucatán
  - Kohler and Milstein Research (Site 6013), Avenida Colón 197, García Ginerés, Mérida, Yucatán
- Philippines (3):
  - De La Salle Health Sciences Institute (Site 9504), Gov. Mangubat Avenue, Cavite City, Cavite
  - Makati Medical Center (Site 9502), No. 2 Amorsolo Street, Legaspi Village, Makati City, National Capital Region
  - Asian Hospital and Medical Center (Site 9503), 2205 Civic Drive, Muntinlupa, National Capital Region
- Puerto Rico AIDS Clinical Trials Unit (Site 1024), Proyecto ACTU Biomedical Building II, San Juan, Puerto Rico
- South Africa (16):
  - Peermed Clinical Trial Center (Site 9215), Corner of Voortrekker and Monument Roads, Kempton Park, Ekurhuleni, Gauteng
  - Worthwhile Clinical Trials (Site 9214), No. 1 Mowbray Avenue, Benoni, Gauteng
  - The Aurum Institute Tembisa Clinical Research Site (Site 9217), Cnr Flint Mazibuko / Rev RTJ Namane Drive, Johannesburg, Gauteng
  - Roodepoort Medicross (Site 9220), 54 Ontdekkers Road, Johannesburg, Gauteng
  - Soweto ACTG CRS (Site 9203), Chris Hani Road, Johannesburg, Gauteng
  - Helen Joseph Hospital (Site 9201), Perth Road, Johannesburg, Gauteng
  - Setshaba Research Centre (Site 9205), 2088 Block H, Pretoria, Gauteng
  - Into Research (Site 9210), Totius Street, Pretoria, Gauteng
  - Durban International Clinical Research Site (Site 9208), Sidmouth Avenue, Durban, KwaZulu-Natal
  - Welkom Clinical Trial Centre (Site 9211), 189 Power Road, Welkom, Matjhabeng, Free State
  - The Aurum Institute Klerksdorp Clinical Research Center (Site 9204), Corner Margaretha Prinsloo St. and O.R. Tambo St., Klerksdorp, North West
  - The Aurum Institute Rustenburg Clinical Research Site (Site 9202), 50 Steen St., c/o Pretorius St., Rustenburg, North West
  - TASK Eden (Site 9218), G, 4 Victoria St., George
  - CLINRESCO, ARWYP Medical Suites (Site 9209), 22 Pine Avenue, Johannesburg
  - Mzansi Ethical Research Centre (Site 9212), 184 Cowen Ntuli Street, Steve Tschwete, Mpumalanga
  - Global Clinical Trials Sunnyside (Site 9216), 175 Steve Biko Street, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data are available from ACTIV-2 clinical trial in accessclinicaldata@NIAID, a NIAID cloud-based secure controlled access data platform that enables sharing of and access to data sets from clinical trials for basic and clinical research and requires a data access request and a signed data use agreement.
Supporting Information: Study Protocol, ICF
Access Criteria: NIAID OCICB requires a Data Use Agreement be signed by investigators seeking to obtain the PUD.
URL: https://accessclinicaldata.niaid.nih.gov/study-viewer/clinical_trials

REFERENCES:
- [Background] Currier JS, Moser C, Eron JJ, Chew KW, Smith DM, Javan AC, Wohl DA, Daar ES, Hughes MD; ACTIV-2/A5401 Study Team. ACTIV-2: A Platform Trial for the Evaluation of Novel Therapeutics for the Treatment of Early COVID-19 in Outpatients. J Infect Dis. 2023 Aug 31;228(Suppl 2):S77-S82. doi: 10.1093/infdis/jiad246. PMID 37650231
- [Background] Chew KW, Moser C, Yeh E, Wohl DA, Daar ES, Ritz J, Javan AC, Eron JJ, Currier JS, Smith DM, Hughes MD; ACTIV-2/A5401 Study Team. Validity and Characterization of Time to Symptom Resolution Outcome Measures in the ACTIV-2/A5401 Outpatient COVID-19 Treatment Trial. J Infect Dis. 2023 Aug 31;228(Suppl 2):S83-S91. doi: 10.1093/infdis/jiad300. PMID 37650237
- [Background] Moser CB, Chew KW, Ritz J, Newell M, Javan AC, Eron JJ, Daar ES, Wohl DA, Currier JS, Smith DM, Hughes MD; ACTIV-2/A5401 Study Team. Pooling Different Placebos as a Control Group in a Randomized Platform Trial: Benefits and Challenges From Experience in the ACTIV-2 COVID-19 Trial. J Infect Dis. 2023 Aug 31;228(Suppl 2):S92-S100. doi: 10.1093/infdis/jiad209. PMID 37650234
- [Background] Moser CB, Chew KW, Giganti MJ, Li JZ, Aga E, Ritz J, Greninger AL, Javan AC, Bender Ignacio R, Daar ES, Wohl DA, Currier JS, Eron JJ, Smith DM, Hughes MD; ACTIV-2/A5401 Study Team. Statistical Challenges When Analyzing SARS-CoV-2 RNA Measurements Below the Assay Limit of Quantification in COVID-19 Clinical Trials. J Infect Dis. 2023 Aug 31;228(Suppl 2):S101-S110. doi: 10.1093/infdis/jiad285. PMID 37650235
- [Result] Bender Ignacio RA, Wohl DA, Arends R, Pilla Reddy V, Mu Y, Javan AC, Hughes MD, Eron JJ, Currier JS, Smith D, Chew KW, Gibbs M, Fletcher CV. Comparative Pharmacokinetics of Tixagevimab/Cilgavimab (AZD7442) Administered Intravenously Versus Intramuscularly in Symptomatic SARS-CoV-2 Infection. Clin Pharmacol Ther. 2022 Dec;112(6):1207-1213. doi: 10.1002/cpt.2706. Epub 2022 Jul 26. PMID 35797235
- [Result] Boucau J, Chew KW, Choudhary MC, Deo R, Regan J, Flynn JP, Crain CR, Hughes MD, Ritz J, Moser C, Dragavon JA, Javan AC, Nirula A, Klekotka P, Greninger AL, Coombs RW, Fischer WA 2nd, Daar ES, Wohl DA, Eron JJ, Currier JS, Smith DM; POSITIVES study team; Li JZ, Barczak AK; ACTIV-2/A5401 Study Team. Monoclonal antibody treatment drives rapid culture conversion in SARS-CoV-2 infection. Cell Rep Med. 2022 Jul 19;3(7):100678. doi: 10.1016/j.xcrm.2022.100678. Epub 2022 Jun 20. PMID 35793677
- [Result] Chew KW, Moser C, Daar ES, Wohl DA, Li JZ, Coombs RW, Ritz J, Giganti M, Javan AC, Li Y, Choudhary MC, Deo R, Malvestutto C, Klekotka P, Price K, Nirula A, Fischer W, Bala V, Ribeiro RM, Perelson AS, Fletcher CV, Eron JJ, Currier JS; ACTIV-2/A5401 Study Team; Hughes MD, Smith DM. Antiviral and clinical activity of bamlanivimab in a randomized trial of non-hospitalized adults with COVID-19. Nat Commun. 2022 Aug 22;13(1):4931. doi: 10.1038/s41467-022-32551-2. PMID 35995785
- [Result] Li Y, Harrison LJ, Chew KW, Currier JS, Wohl DA, Daar ES, Evering TH, Wu R, Giganti M, Ritz J, Javan AC, Coombs RW, Moser C, Hughes MD, Eron JJ, Smith DM, Li JZ. Nasal and Plasma Severe Acute Respiratory Syndrome Coronavirus 2 RNA Levels Are Associated With Timing of Symptom Resolution in the ACTIV-2 Trial of Nonhospitalized Adults With Coronavirus Disease 2019. Clin Infect Dis. 2023 Feb 18;76(4):734-737. doi: 10.1093/cid/ciac818. PMID 36210483
- [Result] Smith DM, Li JZ, Moser C, Yeh E, Currier JS, Chew KW, Hughes MD; ACTIV-2/A5401 Study Team. Recurrence of Symptoms Following a 2-Day Symptom Free Period in Patients With COVID-19. JAMA Netw Open. 2022 Oct 3;5(10):e2238867. doi: 10.1001/jamanetworkopen.2022.38867. PMID 36301549
- [Result] Choudhary MC, Chew KW, Deo R, Flynn JP, Regan J, Crain CR, Moser C, Hughes MD, Ritz J, Ribeiro RM, Ke R, Dragavon JA, Javan AC, Nirula A, Klekotka P, Greninger AL, Fletcher CV, Daar ES, Wohl DA, Eron JJ, Currier JS, Parikh UM, Sieg SF, Perelson AS, Coombs RW, Smith DM, Li JZ; ACTIV-2/A5401 Study Team. Emergence of SARS-CoV-2 escape mutations during Bamlanivimab therapy in a phase II randomized clinical trial. Nat Microbiol. 2022 Nov;7(11):1906-1917. doi: 10.1038/s41564-022-01254-1. Epub 2022 Oct 26. PMID 36289399
- [Result] Moser C, Li JZ, Eron JJ, Aga E, Daar ES, Wohl DA, Coombs RW, Javan AC, Bender Ignacio RA, Jagannathan P, Ritz J, Sieg SF, Parikh UM, Hughes MD, Currier JS, Smith DM, Chew KW; ACTIV-2/A5401 Study Team. Predictors of SARS-CoV-2 RNA From Nasopharyngeal Swabs and Concordance With Other Compartments in Nonhospitalized Adults With Mild to Moderate COVID-19. Open Forum Infect Dis. 2022 Nov 11;9(11):ofac618. doi: 10.1093/ofid/ofac618. eCollection 2022 Nov. PMID 36467293
- [Result] Ramirez SI, Grifoni A, Weiskopf D, Parikh UM, Heaps A, Faraji F, Sieg SF, Ritz J, Moser C, Eron JJ, Currier JS, Klekotka P, Sette A, Wohl DA, Daar ES, Hughes MD, Chew KW, Smith DM, Crotty S; Accelerating COVID-19 Therapeutic Interventions and Vaccines-2/A5401 (ACTIV-2/A5401) Study Team. Bamlanivimab therapy for acute COVID-19 does not blunt SARS-CoV-2-specific memory T cell responses. JCI Insight. 2022 Dec 22;7(24):e163471. doi: 10.1172/jci.insight.163471. PMID 36378539
- [Result] Jilg N, Chew KW, Giganti MJ, Daar ES, Wohl DA, Javan AC, Kantor A, Moser C, Coombs RW, Neytman G, Hoover K, Jana A, Hart PA, Greninger AL, Szurgot B, Eron JJ, Currier JS, Hughes MD, Smith DM, Li JZ; ACTIV-2/A5401 Study Team. One Week of Oral Camostat Versus Placebo in Nonhospitalized Adults With Mild-to-Moderate Coronavirus Disease 2019: A Randomized Controlled Phase 2 Trial. Clin Infect Dis. 2023 Oct 5;77(7):941-949. doi: 10.1093/cid/ciad342. PMID 37279602
- [Result] Taiwo BO, Chew KW, Moser C, Wohl DA, Daar ES, Li JZ, Greninger AL, Bausch C, Luke T, Hoover K, Neytman G, Giganti MJ, Olefsky M, Javan AC, Fletcher CV, Eron JJ, Currier JS, Hughes MD, Smith DM; ACTIV-2/A5401 Study Team. Phase 2 Safety and Antiviral Activity of SAB-185, a Novel Polyclonal Antibody Therapy for Nonhospitalized Adults With COVID-19. J Infect Dis. 2023 Jul 14;228(2):133-142. doi: 10.1093/infdis/jiad013. PMID 36661240
- [Result] Evering TH, Chew KW, Giganti MJ, Moser C, Pinilla M, Wohl DA, Currier JS, Eron JJ, Javan AC, Bender Ignacio R, Margolis D, Zhu Q, Ma J, Zhong L, Yan L, D'Andrea Nores U, Hoover K, Mocherla B, Choudhary MC, Deo R, Ritz J, Fischer WA, Fletcher CV, Li JZ, Hughes MD, Smith D, Daar ES; ACTIV-2/A5401 Study Team. Safety and Efficacy of Combination SARS-CoV-2 Neutralizing Monoclonal Antibodies Amubarvimab Plus Romlusevimab in Nonhospitalized Patients With COVID-19. Ann Intern Med. 2023 May;176(5):658-666. doi: 10.7326/M22-3428. Epub 2023 Apr 18. PMID 37068272
- [Result] Bender Ignacio RA, Chew KW, Moser C, Currier JS, Eron JJ, Javan AC, Giganti MJ, Aga E, Gibbs M, Tchouakam Kouekam H, Johnsson E, Esser MT, Hoover K, Neytman G, Newell M, Daar ES, Fischer W, Fletcher CV, Li JZ, Greninger AL, Coombs RW, Hughes MD, Smith D, Wohl DA; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-2/A5401 Study Team. Safety and Efficacy of Combined Tixagevimab and Cilgavimab Administered Intramuscularly or Intravenously in Nonhospitalized Patients With COVID-19: 2 Randomized Clinical Trials. JAMA Netw Open. 2023 Apr 3;6(4):e2310039. doi: 10.1001/jamanetworkopen.2023.10039. PMID 37099295
- [Result] Deo R, Choudhary MC, Moser C, Ritz J, Daar ES, Wohl DA, Greninger AL, Eron JJ, Currier JS, Hughes MD, Smith DM, Chew KW, Li JZ; ACTIV-2/A5401 Study Team. Symptom and Viral Rebound in Untreated SARS-CoV-2 Infection. Ann Intern Med. 2023 Mar;176(3):348-354. doi: 10.7326/M22-2381. Epub 2023 Feb 21. PMID 36802755
- [Result] Li Y, Moser C, Aga E, Currier JS, Wohl DA, Daar ES, Ritz J, Greninger AL, Sieg S, Parikh UM, Coombs RW, Hughes MD, Eron JJ, Smith DM, Chew KW, Li JZ; ACTIV-2/A5401 Study Team. Immune Status and SARS-CoV-2 Viral Dynamics. J Infect Dis. 2023 Aug 31;228(Suppl 2):S111-S116. doi: 10.1093/infdis/jiad200. PMID 37650232
- [Result] Giganti MJ, Chew KW, Eron JJ, Li JZ, Pinilla M, Moser C, Javan AC, Fischer WA, Klekotka P, Margolis D, Wohl DA, Coombs RW, Daar ES, Smith DM, Currier JS, Hughes MD; ACTIV-2/A5401 Study Team. Association Between Anterior Nasal and Plasma SARS-CoV-2 RNA Levels and Hospitalization or Death in Nonhospitalized Adults With Mild-to-Moderate COVID-19. J Infect Dis. 2023 Aug 31;228(Suppl 2):S117-S125. doi: 10.1093/infdis/jiad287. PMID 37650230
- [Result] Evering TH, Moser CB, Jilg N, Yeh E, Sanusi B, Wohl DA, Daar ES, Li JZ, Klekotka P, Javan AC, Eron JJ, Currier JS, Hughes MD, Smith DM, Chew KW; ACTIV-2/A5401 Study Team. Long COVID After Bamlanivimab Treatment. J Infect Dis. 2023 Aug 31;228(Suppl 2):S126-S135. doi: 10.1093/infdis/jiad286. PMID 37650236
- [Result] Ribeiro RM, Choudhary MC, Deo R, Giganti MJ, Moser C, Ritz J, Greninger AL, Regan J, Flynn JP, Wohl DA, Currier JS, Eron JJ, Hughes MD, Smith DM, Chew KW, Daar ES, Perelson AS, Li JZ; ACTIV-2/A5401 Study Team. Variant-Specific Viral Kinetics in Acute COVID-19. J Infect Dis. 2023 Aug 31;228(Suppl 2):S136-S143. doi: 10.1093/infdis/jiad314. PMID 37650233
- [Result] Kara W. Chew, Carlee B. Moser, Eric S. Daar, David A. Wohl, Eunice Yeh, Justin Ritz, Arzhang Cyrus Javan, Joseph J. Eron, Judith S. Currier, Davey M. Smith, Michael D. Hughes, for the ACTIV-2/A5401 Study Team. SYMPTOM OUTCOME MEASURES FOR OUTPATIENT COVID-19 PHASE 3 TREATMENT TRIALS. Presented at conference, 03/10/2021. 2021 Conference on Retroviruses and Opportunistic Infections (CROI 2021, Chicago, IL and/or Virtual, 03/06/2021 - 03/10/2021. (A5401)
- [Result] Kara W. Chew, Carlee B. Moser, Jonathan Z. Li, Robert W. Coombs, Eric S. Daar, David A. Wohl, Evgenia Aga, Justin Ritz, Arzhang Cyrus Javan, Joseph J. Eron, Judith S. Currier, Michael D. Hughes, Davey M. Smith, for the ACTIV-2/A5401 Study Team. SARS-CoV-2 RNA LEVELS CORRELATE WITH SYMPTOM DURATION BUT NOT SEVERITY IN OUTPATIENTS. Presented at conference, 03/10/2021. 2021 Conference on Retroviruses and Opportunistic Infections (CROI 2021, Chicago, IL and/or Virtual, 03/06/2021 - 03/10/2021. (A5401)
- [Result] Teresa H. Evering, Mark J. Giganti, Kara W. Chew, Michael D. Hughes, Carlee B. Moser, David A. Wohl, Judith S. Currier, Joseph J. Eron, Arzhang Cyrus Javan, David Margolis, Qing Zhu, Ulises D'Andrea, Keila Hoover, Bharat R. Mocherla, Courtney Fletcher, Jonathan Li, Davey M. Smith, Eric S. Daar. SAFETY AND EFFICACY OF COMBINATION SARS-CoV-2 MONOCLONAL NEUTRALIZING ANTIBODIES (MAB) BRII-196 AND BRII-198 IN NON-HOSPITALIZED COVID-19 PATIENTS. Presented at conference, 09/30/2021. 2021 IDWeek, Virtual, 09/20/2021 - 10/03/2021
- [Result] Teresa H. Evering, Busola Sanusi, Nikolaus Jilg, Eunice Yeh, Carlee B. Moser, Justin Ritz, David A. Wohl, Eric S. Daar, Paul Klekotka, Arzhang Cyrus Javan, Joseph J. Eron, Judith S. Currier, Michael D. Hughes, Davey M. Smith, and Kara W. Chew, on behalf of the ACTIV-2/A5401 Study Team and Investigators. PREVALENCE AND CHARACTERISTICS OF POST-ACUTE SEQUELAE OF SARS¬-CoV¬-2 (PASC) IN NON¬-HOSPITALIZED PERSONS WITH COVID-¬19 ENROLLED IN A CLINICAL TRIAL OF EARLY TREATMENT (ACTIV-2). Presented at conference, 12/06/2021. 2021 International Workshop on Long-term Complications of HIV and SARS-¬CoV-¬2, Virtual, 12/06/2021 - 12/09/2021. (A5401)
- [Result] Nikolaus Jilg, Kara W. Chew, Mark J. Giganti, Eric S. Daar, David A. Wohl, Arzhang Cyrus Javan, Amy Kantor, Atasi Jana, Philip A. Hart, Joseph J. Eron, Judith S. Currier, Michael Hughes, Davey M. Smith, Jonathan Z. Li. CAMOSTAT IS NOT EFFECTIVE FOR MILD-MODERATE COVID-19 IN A PHASE 2 TRIAL OF ACTIV-2. Accepted by conference - oral presentation, 01/20/2022. 2022 Conference on Retroviruses and Opportunistic Infections (CROI 2022), Denver, CO, 02/13/2022 - 02/16/2022. (A5401)
- [Result] Babafemi O. Taiwo, Kara W. Chew, Mark Giganti, David A. Wohl, Eric S. Daar, Maxine Olefsky, Rick Finnegan, Jake Miles, Arzhang Cyrus Javan, Jonathan Li, Judith S. Currier, Joseph J. Eron, Michael D. Hughes, Davey M. Smith. PHASE-2 EVALUATION OF SAB-185, A POLYCLONAL ANTIBODY TREATMENT FOR COVID-19 IN ACTIV-2. Accepted by conference - poster presentation, 01/20/2022. 2022 Conference on Retroviruses and Opportunistic Infections (CROI 2022), Denver, CO, 02/13/2022 - 02/16/2022. (A5401)
- [Result] Teresa H. Evering, Busola Sanusi, Nikolaus Jilg, Eunice Yeh, Carlee B. Moser, David A. Wohl, Eric S. Daar, Paul Klekotka, Arzhang Cyrus Javan, Joseph J. Eron, Judith S. Currier, Michael D. Hughes, Davey M. Smith, Kara W. Chew. POST-ACUTE SEQUELAE OF SARS-¬CoV-¬2 IN NON-¬HOSPITALIZED ACTIV-¬2 TRIAL PARTICIPANTS. Accepted by conference - poster presentation, 12/10/2021. 2022 Conference on Retroviruses and Opportunistic Infections (CROI 2022), Denver, CO, 02/13/2022 - 02/16/2022. (A5401)
- [Result] Mark J. Giganti, Kara W. Chew, Joseph J. Eron, Jonathan Z. Li, Mauricio Pinilla, Carlee B. Moser, Arzhang Cyrus Javan, William A. Fischer, Paul Klekotka, David Margolis, David A. Wohl, Robert W. Coombs, Eric S. Daar, Davey M. Smith, Michael D. Hughes, Judith S. Currier, for the ACTIV-2/A5401 Study Team. ASSOCIATION BETWEEN ANTERIOR NASAL AND PLASMA SARS-CoV-2 RNA LEVELS AND HOSPITALIZATION OR DEATH FOR NON-HOSPITALIZED ADULTS WITH MILD-TO-MODERATE COVID-19. Accepted by Conference, 06/30/2022. 2022 IDWeek, Washington DC, 10/19/2022 - 10/23/2022. (A5401)
- [Result] Carlee B. Moser, Jonathan Z. Li, Joseph J. Eron, Evgenia Aga, Eric S. Daar, David A. Wohl, Robert W. Coombs, Arzhang Cyrus Javan, Rachel A Bender Ignacio, Prasanna Jagannathan, Justin Ritz, Scott Sieg, Urvi M. Parikh, Michael D. Hughes, Judith S. Currier, Davey M. Smith, Kara W. Chew. FEMALE SEX AND SARS-CoV-2 SEROSTATUS PREDICT NASOPHARYNGEAL RNA CLEARANCE DURING EARLY COVID-19. Accepted by conference - poster presentation, 09/13/2022. 2022 IDWeek, Washington DC, 10/19/2022 - 10/23/2022. (A5401)
- [Result] Yijia Li, Linda J. Harrison, Kara W. Chew, Joseph J. Eron, Eric S. Daar, David A. Wohl, Ryan Wu, Carlee B. Moser, Justin Ritz, Arzhang Cyrus Javan, Robert W. Coombs, Michael D. Hughes, Judith S. Currier, Davey M. Smith, Jonathan Z. Li. NASAL AND PLASMA SARS-CoV-2 RNA LEVELS PREDICT TIMING OF SYMPTOM RESOLUTION IN THE ACTIV-2 TRIAL OF NON-HOSPITALIZED ADULTS WITH COVID-19. Accepted by conference - oral presentation, 09/12/2022. 2022 IDWeek, Washington DC, 10/19/2022 - 10/23/2022. (A5401)
- [Result] Teresa H. Evering*, Carlee B. Moser*, Nikolaus Jilg, Justin Ritz, David A. Wohl, Jonathan Z. Li, David Margolis, Arzhang Cyrus Javan, Joseph J. Eron, Judith S. Currier, Eric S. Daar, Davey M. Smith*, Michael D. Hughes*, Kara W. Chew*, for the ACTIV-2/A5401 Study Team. *Contributed equally. POST-ACUTE COVID OUTCOMES: AMUBARVIMAB+ROMLUSEVIMAB VS PLACEBO IN THE ACTIV-2 TRIAL. Accepted by conference - poster presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. Submitted for Review, 12/08/2022. (A5401).
- [Result] Yijia Li, Carlee B. Moser, Evgenia Aga, Judith S. Currier, David A. Wohl, Eric S. Daar, Justin Ritz, Robert W. Coombs, Michael D. Hughes, Joseph J. Eron, Davey M. Smith, Kara W. Chew, Jonathan Z. Li. IMMUNE STATUS AND SARS-COV-2 VIRAL DYNAMICS. Accepted by conference - poster presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Rinki Deo, Manish C. Choudhary, Carlee B. Moser, Justin Ritz, Eric S. Daar, David A. Wohl, Alexander L. Greninger, Joseph J. Eron, Judith S. Currier, Michael D. Hughes*, Davey M. Smith*, Kara W. Chew*, Jonathan Z. Li*, for the ACTIV-2/A5401 Study Team. *Contributed equally. SYMPTOM AND VIRAL REBOUND IN UNTREATED COVID-19 INFECTION. Accepted by conference - oral presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Rachel Bender Ignacio*, Kara W. Chew*, Carlee B. Moser, Judith S. Currier, Joseph J. Eron, Arzhang Cyrus Javan, Evgenia Aga, Michael Gibbs, Herve Tchouakam Kouekam, Matthew Newell, Eric S. Daar, Jonathan Z. Li, Michael D. Hughes, Davey M. Smith, and David A. Wohl, for the ACTIV-2/A5401 Study Team. TIXAGEVIMAB/CILGAVIMAB IM AND IV IN SYMPTOMATIC COVID-19: A RANDOMIZED CONTROLLED ACTIV-2 TRIAL. Accepted by conference - poster presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Nikolaus Jilg, Mark J. Giganti, Kara W. Chew, Kathryn Shaw-Saliba, Justin Ritz, Carlee B. Moser, Teresa H. Evering, Eric S. Daar, Joseph J. Eron, Judith S. Currier, Michael D. Hughes, H. Cliff Lane, Robin L. Dewar*, Davey M. Smith*, Jonathan Z. Li*. *Contributed equally. PLASMA ANTIBODY AND N ANTIGEN STATUS PREDICT OUTCOMES IN OUTPATIENTS WITH COVID-19. Accepted by conference - poster presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Prasanna Jagannathan*, Kara W. Chew*, Mark J. Giganti, Michael D. Hughes, Mark Main, Phillip Monk, Arzhang Cyrus Javan, Jonathan Z. Li, David A. Wohl, Eric S. Daar, Joseph J. Eron, Judith S. Currier, Upinder Singh*, Davey M. Smith*, William Fischer*. *Contributed equally. SAFETY AND EFFICACY OF INHALED INTERFERON-β1A (SNG001) IN OUTPATIENTS WITH COVID-19. Accepted by conference - oral presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Manish C. Choudhary, Rinki Deo, Teresa H. Evering, Kara W. Chew, Mark J. Giganti, Carlee B. Moser, Justin Ritz, David A. Wohl, Judith S. Currier, Joseph J. Eron, David Margolis, Yun Ji, Michael D. Hughes, Davey M. Smith, Eric S. Daar, Jonathan Z. Li for the ACTIV-2/A5401 Study Team. CHARACTERIZATION OF SINGLE VERSUS DUAL ACTIVE MONOCLONAL ANTIBODIES AGAINST SARS-CoV-2. Accepted by conference - oral presentation. 2023 30th Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 02/19/2023 - 02/22/2023. (A5401)
- [Result] Jagannathan P, Chew KW, Giganti MJ, Hughes MD, Moser C, Main MJ, Monk PD, Javan AC, Li JZ, Fletcher CV, McCarthy C, Wohl DA, Daar ES, Eron JJ, Currier JS, Singh U, Smith DM, Fischer W; ACTIV-2/A5401 Study Team. Safety and efficacy of inhaled interferon-beta1a (SNG001) in adults with mild-to-moderate COVID-19: a randomized, controlled, phase II trial. EClinicalMedicine. 2023 Oct 6;65:102250. doi: 10.1016/j.eclinm.2023.102250. eCollection 2023 Nov. PMID 37855026
- [Derived] Chew KW, Taiwo BO, Moser C, Daar ES, Wohl DA, Ritz J, Javan AC, Li JZ, Fischer W, Greninger AL, Bausch C, Luke T, Call R, Neytman G, Giganti MJ, Fletcher CV, Hughes MD, Eron JJ, Currier JS, Smith DM; ACTIV-2/A5401 Study Team. Safety and Efficacy of SAB-185 for Nonhospitalized Adults With COVID-19: A Randomized Clinical Trial. J Infect Dis. 2024 Nov 15;230(5):1177-1186. doi: 10.1093/infdis/jiae369. PMID 39028902
- [Derived] Jilg N, Giganti MJ, Chew KW, Shaw-Saliba K, Ritz J, Moser C, Evering TH, Daar ES, Eron JJ, Currier JS, Hughes MD, Lane HC, Dewar R, Smith DM, Li JZ. SARS-CoV-2 Plasma Antibody and Nucleocapsid Antigen Status Predict Outcomes in Outpatients With COVID-19. Clin Infect Dis. 2024 Oct 15;79(4):920-927. doi: 10.1093/cid/ciae324. PMID 39018444
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Chew KW, Moser C, Daar ES, Wohl DA, Li JZ, Coombs R, Ritz J, Giganti M, Javan AC, Li Y, Malvestutto C, Klekotka P, Price K, Nirula A, Fischer W, Bala V, Ribeiro RM, Perelson AS, Fletcher CV, Eron JJ, Currier JS, Hughes MD, Smith DM; ACTIV-2/A5401 Study Team. Bamlanivimab reduces nasopharyngeal SARS-CoV-2 RNA levels but not symptom duration in non-hospitalized adults with COVID-19: A Phase 2 Randomized Clinical Trial. medRxiv [Preprint]. 2021 Dec 21:2021.12.17.21268009. doi: 10.1101/2021.12.17.21268009. PMID 34981077
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — https://www.cdc.gov/coronavirus/2019-nCoV/index.html
- See also: A Participant's Guide to Clinical Trials (NIAID) — https://www.niaid.nih.gov/clinical-trials/participant-guide
- See also: Find a Clinical Trial (NIAID) — https://www.niaid.nih.gov/clinical-trials/find-a-clinical-trial
- See also: Clinical Trials at NIAID — https://www.niaid.nih.gov/clinical-trials
- See also: National Institute for Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: WHO COVID-19 treatment guidelines — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were considered to be separately enrolled participants for subsequent phases of the study.
  BRII arms included pooled participants from Phase 2/Phase 3 to complete a Phase 3 analysis.
Groups:
- AZD7442 (IV) Placebo (Phase 2): Administered by IV infusion.
  Placebo for AZD7442 (IV): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- AZD7442 (IM) Placebo (Phase 2): Administered by IM injection.
  Placebo for AZD7442 (IM): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- SNG001 Placebo (Phase 2): Administered by inhalation.
  Placebo for SNG001: Trisodium citrate dihydrate, di-sodium hydrogen-phosphate, sodium dihydrogen-phosphate dihydrate, racemic methionine (DL-methionine) and water. 1.3 mL solution administered once daily for 14 days using Aerogen Ultra nebulizer (inhalation device). Participants are no longer being randomized to this intervention.
- Camostat Pooled Placebo (Phase 2): Administered as oral tablets.
  Placebo for Camostat: 200 mg (2 x 100 mg) film-coated tablets administered orally every 6 hours for 7 days. Participants are no longer being randomized to this intervention.
- SAB-185 (Low Dose) Placebo (Phase 2): Administered by IV infusion.
  Placebo for SAB-185 (low dose): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- SAB-185 (Low Dose) (Phase 3) OMICRON Population: Administered by IV infusion.
  SAB-185 (3,840 Units/kg): Administered by IV infusion as a single dose. Participants are no longer being randomized to this intervention.
  The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- Casirivimab and Imdevimab (Phase 3) OMICRON Population: Administered by IV infusion.
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as a single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
  The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population: Administered by IV infusion
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population: Administered by IV infusion
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- SAB-185 (High Dose) Placebo (Phase 2): Administered by IV infusion.
  Placebo for SAB-185 (high dose): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- BMS 986414+BMS 986413 Placebo (Phase 2): Administered as subcutaneous (SC) injections.
  Placebo for BMS-986414 + BMS-986413: Administered SC as 4 separate injections for one dose. Participants are no longer being randomized to this intervention.
Period: Overall Study
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Placebo (Phase 2)
Started (Total enrolled = Started (Randomized) + Screen Fail (Randomized) + Excluded from Analysis at NIH Request (suspected scientific misconduct at site level) + Dual Enrolled Subject = 3923+2+118+1=4044 A*= Subjects Treated and then not completed for reported reason and not excluded from analyses = 0 + 325 + 204 + 36 + 31 + 38 + 1 = 635 Not completed=A*+Ongoing+Randomized not Treated+Screen failed but randomized+Excluded from Analyses+Dual Enrolled Subject = 635 + 0 + 54 + 2 + 252 +1) | 48 | 46 | 111 | 114 | 1079 | 424 | 422 | 61 | 33 | 110 | 54 | 110 | 53 | 113 | 54 | 110 | 39 | 225 | 214 | 142 | 153 | 115 | 41 | 112 | 61
Completed | 45 | 43 | 100 | 101 | 843 | 329 | 328 | 42 | 23 | 77 | 36 | 88 | 41 | 79 | 38 | 84 | 26 | 167 | 156 | 102 | 110 | 81 | 35 | 84 | 42
Not Completed | 3 | 3 | 11 | 13 | 236 | 95 | 94 | 19 | 10 | 33 | 18 | 22 | 12 | 34 | 16 | 26 | 13 | 58 | 58 | 40 | 43 | 34 | 6 | 28 | 19
Not completed — Lost to Follow-up | 1 | 1 | 8 | 5 | 92 | 25 | 25 | 3 | 2 | 13 | 9 | 13 | 9 | 13 | 8 | 10 | 6 | 13 | 21 | 6 | 7 | 21 | 1 | 7 | 6
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3 | 20 | 20 | 25 | 6 | 1 | 12 | 5 | 7 | 2 | 13 | 4 | 9 | 0 | 15 | 12 | 9 | 14 | 3 | 2 | 9 | 8
Not completed — Other | 1 | 0 | 0 | 1 | 6 | 6 | 5 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 17 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 12 | 2 | 11 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Requirement to start alternative therapy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 2 | 6 | 4 | 3 | 3 | 0 | 4 | 0 | 0 | 1 | 3 | 3 | 3 | 4 | 5 | 4 | 0 | 0 | 5 | 0 | 3 | 1
Not completed — Screen Fail but Randomized | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Excluded from analysis at NIH request (due to suspected scientific misconduct at site level) | 0 | 0 | 0 | 0 | 81 | 37 | 23 | 4 | 6 | 3 | 4 | 0 | 0 | 4 | 0 | 1 | 1 | 21 | 16 | 21 | 19 | 3 | 2 | 4 | 2
Not completed — Dual Enrolled Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total MITT Population=Randomized and Treated and included in analysis = All with Randomization Date - Randomized Not Treated-Randomized screen failed - Excluded from analysis - Dual enrollment = 4044 - 54 - 2 - 252 - 1
  All participants were considered to be separately enrolled participants for subsequent phases of the study.
  BRII arms included pooled participants from Phase 2/Phase 3 to complete a Phase 3 analysis.
Groups:
- Camostat Placebo (Phase 2): Administered as oral tablets.
  Placebo for Camostat: 200 mg (2 x 100 mg) film-coated tablets administered orally every 6 hours for 7 days. Participants are no longer being randomized to this intervention.
- SAB-185 (Low Dose) (Phase 3) OMICRON Population: Administered by IV infusion.
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- Casirivimab and Imdevimab (Phase 3) OMICRON Population: Administered by IV infusion
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
  The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
- Total: Total of all reporting groups
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Placebo (Phase 2) | Camostat (Phase 2) | Camostat Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) NON-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Placebo (Phase 2) | Total
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 990 | 383 | 396 | 54 | 27 | 103 | 50 | 110 | 52 | 106 | 51 | 106 | 34 | 198 | 194 | 121 | 134 | 107 | 39 | 105 | 58 | 3735
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (15.80) | 41.5 (13.79) | 45.2 (13.52) | 46.7 (13.69) | 51.1 (15.92) | 47.8 (13.59) | 48.7 (13.68) | 42.5 (12.06) | 44.6 (13.63) | 39.9 (11.80) | 36.8 (12.07) | 40.2 (12.37) | 40.1 (12.05) | 37.7 (12.72) | 38.5 (11.57) | 39.0 (10.94) | 37.3 (11.22) | 50.1 (14.23) | 52.8 (15.86) | 54.9 (13.12) | 52.7 (14.16) | 39.9 (12.47) | 40.6 (14.88) | 42.8 (14.57) | 41.4 (13.02) | 47.2 (14.99)
Age, Customized [Count of Participants; unit: Participants]
  Younger than 55 | 30 | 35 | 84 | 81 | 582 | 254 | 256 | 45 | 21 | 92 | 46 | 98 | 44 | 97 | 44 | 100 | 32 | 115 | 105 | 52 | 62 | 92 | 32 | 84 | 48 | 2531
  55 or older | 18 | 11 | 27 | 31 | 408 | 129 | 140 | 9 | 6 | 11 | 4 | 12 | 8 | 9 | 7 | 6 | 2 | 83 | 89 | 69 | 72 | 15 | 7 | 21 | 10 | 1204
  Younger than 60 | 37 | 42 | 98 | 93 | 691 | 302 | 303 | 50 | 22 | 99 | 49 | 106 | 49 | 103 | 48 | 102 | 34 | 146 | 131 | 76 | 93 | 100 | 34 | 90 | 52 | 2950
  60 or older | 11 | 4 | 13 | 19 | 299 | 81 | 93 | 4 | 5 | 4 | 1 | 4 | 3 | 3 | 3 | 4 | 0 | 52 | 63 | 45 | 41 | 7 | 5 | 15 | 6 | 785
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 54 | 56 | 515 | 197 | 209 | 33 | 16 | 51 | 30 | 66 | 26 | 62 | 26 | 62 | 16 | 108 | 107 | 72 | 67 | 59 | 22 | 57 | 29 | 1989
  Male | 22 | 23 | 57 | 56 | 475 | 186 | 187 | 21 | 11 | 52 | 20 | 44 | 26 | 44 | 25 | 44 | 18 | 90 | 87 | 49 | 67 | 48 | 17 | 48 | 29 | 1746
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 18 | 31 | 328 | 190 | 191 | 24 | 13 | 49 | 16 | 58 | 27 | 58 | 27 | 45 | 18 | 117 | 100 | 62 | 55 | 44 | 22 | 54 | 37 | 1616
  Not Hispanic or Latino | 33 | 28 | 93 | 79 | 660 | 193 | 205 | 30 | 14 | 54 | 34 | 52 | 25 | 48 | 24 | 61 | 16 | 81 | 94 | 59 | 79 | 63 | 17 | 51 | 21 | 2114
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 5 | 2 | 4 | 57 | 15 | 22 | 1 | 0 | 2 | 1 | 3 | 3 | 3 | 1 | 4 | 1 | 4 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 134
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 2 | 4 | 1 | 0 | 1 | 0 | 32
  Black or African American | 3 | 2 | 13 | 10 | 63 | 79 | 62 | 9 | 4 | 8 | 8 | 13 | 3 | 4 | 7 | 9 | 1 | 17 | 16 | 4 | 12 | 15 | 1 | 10 | 8 | 381
  Multiple | 3 | 0 | 0 | 2 | 7 | 4 | 2 | 0 | 1 | 2 | 1 | 5 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 34
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
  Other | 1 | 2 | 3 | 3 | 16 | 14 | 15 | 0 | 1 | 4 | 1 | 3 | 5 | 3 | 1 | 2 | 1 | 11 | 10 | 0 | 0 | 1 | 0 | 2 | 1 | 100
  White | 41 | 37 | 92 | 92 | 840 | 270 | 293 | 44 | 21 | 85 | 38 | 85 | 40 | 95 | 42 | 89 | 30 | 156 | 154 | 113 | 117 | 86 | 38 | 90 | 49 | 3037
  Not collected or reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 10
Baseline BMI (kg/m2 ) [Mean (Standard Deviation); unit: kg/m2] — Population: Data missing for 92 participants
  kg/m2
    number analyzed (Participants) | 42 | 39 | 95 | 97 | 961 | 377 | 394 | 53 | 26 | 103 | 50 | 108 | 52 | 105 | 51 | 103 | 33 | 198 | 194 | 121 | 134 | 105 | 39 | 105 | 58 | 3643
    (all) | 28.4 (4.62) | 29.2 (7.20) | 29.7 (6.08) | 28.3 (6.28) | 29.5 (6.81) | 30.7 (7.44) | 31.4 (7.25) | 32.8 (8.70) | 30.3 (7.81) | 28.9 (5.94) | 28.7 (5.47) | 27.9 (6.95) | 27.9 (5.20) | 28.4 (6.26) | 27.4 (4.93) | 28.0 (7.37) | 27.8 (6.01) | 32.9 (7.84) | 33.1 (7.59) | 31.3 (6.49) | 33.7 (7.09) | 28.1 (6.13) | 29.4 (4.44) | 28.0 (5.43) | 27.1 (4.63) | 30.1 (7.03)
BMI category (kg/m2 ) [Count of Participants; unit: Participants]
  Less than or equal to 35 kg/m2 | 38 | 34 | 77 | 86 | 799 | 278 | 279 | 31 | 19 | 89 | 45 | 99 | 48 | 94 | 50 | 95 | 30 | 116 | 117 | 81 | 73 | 92 | 35 | 96 | 56 | 2857
  Greater than 35 kg/m2 | 4 | 5 | 18 | 11 | 162 | 99 | 115 | 22 | 7 | 14 | 5 | 9 | 4 | 11 | 1 | 8 | 3 | 82 | 77 | 40 | 61 | 13 | 4 | 9 | 2 | 786
  Participants with missing data | 6 | 7 | 16 | 15 | 29 | 6 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 92

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Symptom Duration (Phase 2)
Description: Bamlanivimab arms:
  Symptom duration=max. duration (days) across targeted symptoms including: feeling feverish, cough, shortness of breath/difficulty breathing at rest/with activity, sore throat, body pain/muscle pain/aches, fatigue, headache, chills, nasal obstruction/congestion, nasal discharge, nausea, vomiting, and diarrhea. Subjects who die on/before day 28 assigned symptom duration 29 days.
  No scale. Min. value: 0 Days, Max. Value 29 Days. Higher value=worse health condition.
  Non-Bamlanivimab arms:
  13 symptoms (as for Bamlanivimab) scored daily as absent (score 0), mild (score 1), moderate (score 2) or severe (score 3). Symptom duration=time (days) from Day 0 (pre-treatment) to first of two consecutive days when all symptoms scored moderate/severe at Day 0 (pre-treatment) are scored mild/absent, AND all symptoms scored mild/absent at Day 0 (pre-treatment) are scored absent.
  No scale. Min. value: 0 Days, Max. Value 26 Days. Higher value=worse health condition.
Time Frame: Up to Day 28
Population: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  All placebo arms except for Bamlanivimab include pooled placebo data.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Bamlanivimab 7000mg (Phase 2): Administered by IV infusion.
  Bamlanivimab 7000mg: Administered by single IV infusion. Participants are no longer being randomized to this intervention.
- SAB-185 (Low Dose) Pooled Placebo (Phase 2): Administered by IV infusion; includes SAB-185 (high dose) and placebo from other comparator arms in the study.
  Placebo for SAB-185 (low dose): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- SAB-185 (High Dose) Pooled Placebo (Phase 2): Administered by IV infusion; includes SAB-185 (low dose) and placebo from other comparator arms in the study.
  Placebo for SAB-185 (high dose): Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
Arm/Group | Bamlanivimab 7000mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 107 | 102 | 105 | 107
Days | 21.0 [NA to NA] — Lilly agent symptom duration is analyzed differently from other agents and the median reported is descriptive median without associated probability distribution. Hence 95% CI is not applicable here. Inter-Quartile Range 21 is reported instead for Lilly agent arms. | 18.5 [NA to NA] — Lilly agent symptom duration is analyzed differently from other agents and the median reported is descriptive median without associated probability distribution. Hence 95% CI is not applicable here. Inter-Quartile Range 21 is reported instead for Lilly agent arms. | 24.0 [NA to NA] — Lilly agent symptom duration is analyzed differently from other agents and the median reported is descriptive median without associated probability distribution. Hence 95% CI is not applicable here. Inter-Quartile Range 14 is reported instead for Lilly agent arms. | 20.5 [NA to NA] — Lilly agent symptom duration is analyzed differently from other agents and the median reported is descriptive median without associated probability distribution. Hence 95% CI is not applicable here. Inter-Quartile Range 19 is reported instead for Lilly agent arms. | 11.00 [9.00 to 15.00] | 10.00 [7.00 to 15.00] | 8.00 [7.00 to 12.00] | 10.00 [8.00 to 13.00] | 13.0 [10.0 to 16.0] | 9.0 [8.0 to 12.0] | 9 [8 to 12] | 9 [8 to 13] | 11.0 [10.0 to 13.0] | 10.0 [8.0 to 13.0] | 8.0 [7.0 to 10.0] | 10.0 [8.0 to 13.0] | 8.0 [6.00 to 10.00] | 10.0 [8.00 to 13.00]

2. Primary Outcome: Quantification of SARS-CoV-2 RNA (Phase 2)
Description: Bamlanivimab Agent arms:
  Measured as Detected or Undetected from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Detection is 1.4 (log 10 copies/ml).
  Non-Bamlanivimab Agent arms:
  Measured as below Lower Limit of Quantification (LLoQ) or at/above LLoQ from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Quantification is 2 (log 10 copies/ml).
  SNG001 and SNG001 Pooled Placebo arm each exclude 6 participants, due to unsuitable sample specimen conditions.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 46 | 44 | 105 | 107 | 49 | 44 | 83 | 88 | 93 | 94 | 88 | 80 | 83 | 89 | 91 | 88 | 105 | 107
Participants
  Undetected (less than LLOQ) | 8 | 8 | 8 | 7 | 25 | 23 | 26 | 36 | 26 | 37 | 28 | 32 | 39 | 34 | 35 | 32 | 42 | 44
  Detected (greater than or equal to LLOQ) | 38 | 36 | 97 | 100 | 24 | 21 | 57 | 52 | 67 | 57 | 60 | 48 | 44 | 55 | 56 | 56 | 46 | 49
  Participants with missing records or excluded due to unsuitable sample specimen conditions | 2 | 2 | 6 | 5 | 6 | 7 | 20 | 23 | 17 | 16 | 18 | 25 | 23 | 14 | 16 | 14 | 17 | 14

3. Primary Outcome: Quantification of SARS-CoV-2 RNA (Phase 2)
Description: Bamlanivimab Agent arms:
  Measured as Detected or Undetected from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Detection is 1.4 (log 10 copies/ml).
  Non-Bamlanivimab Agent arms:
  Measured as below Lower Limit of Quantification (LLoQ) or at/above LLoQ from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Quantification is 2 (log 10 copies/ml).
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 46 | 43 | 104 | 106 | 47 | 44 | 83 | 93 | 93 | 94 | 84 | 89 | 91 | 83 | 93 | 82 | 105 | 107
Participants
  Undetected (less than LLOQ) | 11 | 10 | 13 | 17 | 35 | 31 | 66 | 59 | 60 | 62 | 53 | 60 | 63 | 54 | 69 | 52 | 71 | 64
  Detected (greater than or equal to LLOQ) | 35 | 33 | 91 | 89 | 12 | 13 | 17 | 34 | 33 | 32 | 31 | 29 | 28 | 29 | 24 | 30 | 19 | 24
  Participants with missing records or excluded due to unsuitable sample specimen conditions | 2 | 3 | 7 | 6 | 8 | 7 | 20 | 18 | 17 | 16 | 22 | 16 | 15 | 20 | 14 | 20 | 15 | 19

4. Primary Outcome: Quantification of SARS-CoV-2 RNA (Phase 2)
Description: as for outcome 3
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 46 | 42 | 100 | 102 | 46 | 45 | 82 | 91 | 94 | 91 | 84 | 85 | 90 | 86 | 91 | 84 | 105 | 107
Participants
  Undetected (less than LLOQ) | 24 | 28 | 35 | 33 | 44 | 42 | 70 | 81 | 85 | 83 | 73 | 75 | 81 | 81 | 85 | 78 | 82 | 85
  Detected (greater than or equal to LLOQ) | 22 | 14 | 65 | 69 | 2 | 3 | 12 | 10 | 9 | 8 | 11 | 10 | 9 | 5 | 6 | 6 | 8 | 7
  Participants with missing records or excluded due to unsuitable sample specimen conditions | 2 | 4 | 11 | 10 | 9 | 6 | 21 | 20 | 16 | 19 | 22 | 20 | 16 | 17 | 16 | 18 | 15 | 15

5. Primary Outcome: Number of Participants With New Adverse Event (AE) ≥ Grade 3 (Phase 2)
Description: AE Severity: Adverse event Severity grading followed Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017, which can be found on the DAIDS RSC website at:
  https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables.
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death
Time Frame: Thru Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 107 | 102 | 105 | 107
Participants | 6 | 6 | 12 | 6 | 4 | 6 | 10 | 8 | 4 | 9 | 10 | 8 | 5 | 11 | 10 | 10 | 6 | 15

6. Primary Outcome: Cumulative Incidence of Death Due to Any Cause or Hospitalization Due to Any Cause (Phase 3)
Description: Hospitalization defined as ≥24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address medical needs of those with severe COVID-19. An event is defined as first occurrence of hospitalization/death (i.e. if subject has multiple hospitalizations, only the first hospitalization is counted as an event). Therefore, an event can only occur once for a subject. Results are presented as number of events.
Time Frame: Thru Day 28
Population: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Number; unit: Events
Groups:
- SAB-185 (Low Dose) (Phase 3) OMICRON Population: Administered by IV infusion
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
  The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 990 | 383 | 397 | 198 | 194 | 121 | 134
Events | 35 | 8 | 44 | 5 | 3 | 6 | 3

7. Primary Outcome: Proportion of Participants With New Adverse Event (AE) ≥ Grade 3 (Phase 3)
Description: as for outcome 5
Time Frame: Thru Day 28
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population: Administered by IV infusion
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
- Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population: Administered by IV infusion
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 990 | 383 | 397 | 198 | 194 | 121 | 134
Participants | 71 | 30 | 67 | 28 | 16 | 17 | 20

8. Secondary Outcome: COVID-19 Symptom Duration (Phase 3)
Description: Bamlanivimab arm:
  Symptom duration=max. duration (days) across targeted symptoms including: feeling feverish, cough, shortness of breath/difficulty breathing at rest/with activity, sore throat, body pain/muscle pain/aches, fatigue, headache, chills, nasal obstruction/congestion, nasal discharge, nausea, vomiting, and diarrhea. Subjects who die on/before day 28 assigned symptom duration 29 days.
  No scale. Min. value: 0 Days, Max. Value 29 Days. Higher value=worse health condition.
  Non-Bamlanivimab arms:
  13 symptoms (as for Bamlanivimab) scored daily as absent (score 0), mild (score 1), moderate (score 2) or severe (score 3). Symptom duration=time (days) from Day 0 (pre-treatment) to first of two consecutive days when all symptoms scored moderate/severe at Day 0 (pre-treatment) are scored mild/absent, AND all symptoms scored mild/absent at Day 0 (pre-treatment) are scored absent.
  No scale. Min. value: 0 Days, Max. Value 26 Days. Higher value=worse health condition.
Time Frame: Thru Day 28
Population: Analysis population description (Phase 3): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 990 | 383 | 397 | 198 | 194 | 121 | 134
Days | 21.5 [NA to NA] — Lilly agent symptom duration is analyzed differently from other agents and the median reported is descriptive median without associated probability distribution. Hence 95% CI is not applicable here. Inter-Quartile Range 18 is reported instead for Lilly agent arms. | 11.0 [10.0 to 12.0] | 11.0 [10.0 to 13.0] | 11.0 [9.0 to 13.0] | 13.00 [10.0 to 15.0] | 11.0 [9.0 to 14.0] | 14.0 [9.0 to 16.0]

9. Secondary Outcome: Quantification of SARS-CoV-2 RNA (Phase 3)
Description: Measured as Detected or Undetected from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Detection is 1.4 (log 10 copies/ml).
  Non-Bamlanivimab Agent arms:
  Measured as below Lower Limit of Quantification (LLoQ) or at/above LLoQ from staff-collected NP (nasopharyngeal) swabs. Lower Limit of Quantification is 2 (log 10 copies/ml).
Time Frame: Day 3
Population: Analysis population description (Phase 3): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject). All placebo arms = pooled placebo data. BRII-196+BRII-198 data is Ph2 subjects only. Bamlanivimab 700mg (Ph3) enrolled under Prot. v1, OM new in v8 so OM not pre-specified, not done. Participants missing records or unsuitable sample specimen conditions excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 0 | 100 | 93 | 166 | 158 | 113 | 120
Participants
  Undetected (less than LLOQ) |  | 37 | 35 | 47 | 47 | 57 | 51
  Detected (greater than or equal to LLOQ) |  | 63 | 58 | 119 | 111 | 56 | 69
  Participants with missing records or excluded due to unsuitable sample specimen conditions |  | 12 | 16 | 32 | 36 | 8 | 14

10. Secondary Outcome: Cumulative Incidence of Death From Any Cause or Hospitalization Due to Any Cause (Phase 2)
Description: as for outcome 6
Time Frame: Thru Day 28
Population: Analysis population description (Phase 2): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  All placebo arms except for Bamlanivimab include pooled placebo data.
Measure: Number; unit: Events
Arm/Group | Bamlanivimab 7000mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 107 | 102 | 105 | 107
Events | 2 | 4 | 4 | 4 | 0 | 4 | 4 | 7 | 1 | 7 | 6 | 5 | 2 | 4 | 5 | 4 | 6 | 4

11. Secondary Outcome: Cumulative Incidence of Death From Any Cause, or Hospitalization Due to Any Cause Related to COVID-19 (Phase 3)
Description: Hospitalizations due to any cause deemed unrelated to COVID-19 are excluded. Hospitalization defined as ≥24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address medical needs of those with severe COVID-19. An event is defined as first occurrence of hospitalization/death (i.e. if subject has multiple hospitalizations, only the first hospitalization is counted as an event). Therefore, an event can only occur once for a subject. Results are presented as number of events.
Time Frame: Thru Day 28
Population: Analysis population description (Phase 3): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Bamlanivimab 700mg (Phase 3) enrolled under Protocol v1, BRII enrolled under v6 or earlier, this OM was a new addition in v8 so this OM was not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Number; unit: Events
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 0 | 0 | 0 | 198 | 194 | 121 | 134
Events |  |  |  | 4 | 3 | 6 | 2

12. Secondary Outcome: Level of SARS-CoV-2 RNA From NP Swabs (Phase 2)
Description: Measured from staff-collected NP swabs
Time Frame: Thru Day 14
Population: Analysis population description (Phase 2): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject). Participants with missing or unsuitable samples were excluded from analysis.
  All placebo arms except for Bamlanivimab include pooled placebo data.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Bamlanivimab 7000mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 46 | 42 | 100 | 102 | 46 | 45 | 82 | 91 | 94 | 91 | 84 | 85 | 90 | 86 | 91 | 84 | 90 | 92
log 10 copies/mL | 1.357 (0.8371) | 1.201 (0.8123) | 1.669 (1.0883) | 1.552 (0.7373) | 1.09 (0.565) | 1.15 (0.655) | 1.20 (0.857) | 1.32 (0.740) | 1.051 (0.6425) | 1.114 (0.6786) | 1.315 (0.7722) | 1.316 (0.7152) | 1.095 (0.8025) | 0.953 (0.5247) | 0.950 (0.6005) | 0.976 (0.5428) | 1.1 (NA) — Standard deviation not calculated by BMS. Interquartile range is 0.70 to 1.70. | 1.0 (NA) — Standard deviation not calculated by BMS. Interquartile range is 0.70 to 0.70.

13. Secondary Outcome: Level of SARS-CoV-2 RNA From NP Swabs (Phase 3)
Description: Measured from staff-collected NP swabs
Time Frame: Day 3
Population: Bamlanivimab 700mg (Phase 3) enrolled under Protocol v1, this OM was a new addition in v7 so this OM was not pre-specified and therefore not done. Participants with missing records or excluded due to unsuitable sample specimen conditions.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population
Number analyzed (Participants) | 0 | 100 | 93 | 166 | 158 | 113 | 120
log 10 copies/mL |  | 2.899 (1.5822) | 3.122 (2.0459) | 3.960 (2.1722) | 3.857 (2.2445) | 2.745 (2.1912) | 2.935 (2.0670)

14. Secondary Outcome: Duration of Targeted Clinical COVID-19 Symptoms (Phases 2 and 3)
Description: Duration defined as the number of days from start of investigational agent to the first of four consecutive days when all symptoms scored as absent. Targeted symptoms are: Feeling feverish; cough, shortness of breath or difficulty breathing; sore throat; body pain or muscle pain/aches; fatigue (low energy); headache, chills, nasal obstruction or congestion (stuffy nose); nasal discharge (runny nose); nausea or vomiting; and diarrhea. Each symptom is scored daily by the participant as absent (score 0), mild (1), moderate (2) or severe (3)
Time Frame: Thru Day 28
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Bamlanivimab Ph2&3 enrolled under v1, Camostat, SNG001, SAB Ph2 enrolled under Protocol v6 or earlier, this OM was a new addition in protocol v8 so this OM was not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population: Administered by IV infusion.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
- Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population: Administered by IV infusion.
  The "Non-Omicron subpopulation" enrolled under Protocol Version 7 was defined as all participants enrolled under Protocol Version 7 excluding those in the "Omicron subpopulation."
  Omicron/Non-Omicron subpopulation definitions were updated in Version 10.0 of the Primary SAP to be based on the timing of emergence of the Omicron variant within the study population as follows:
  * Variant information from any sample (i.e., not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol Version 7.0 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
- SAB-185 (Low Dose) (Phase 3) OMICRON Population: Administered by IV infusion The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  SAB-185 (3,840 Units/kg): Administered by IV infusion as single dose. Participants are no longer being randomized to this intervention.
- Casirivimab and Imdevimab (Phase 3) OMICRON Population: Administered by IV infusion The "Omicron subpopulation" enrolled under Protocol v.7 was defined as (1) all participants randomized under Protocol v.7 infected with the Omicron variant as identified on sequencing of NP sample obtained on day 0, plus (2) all participants randomized under Protocol v.7 on/after December 26, 2021, who do not have variant information available from sample obtained on day 0.
  Definitions were updated in Primary SAP v10.0 to be based on timing of emergence of Omicron variant within the study population as follows:
  * Variant information from any sample (i.e. not just from samples obtained on day 0) could be used to assign a participant to the Omicron or non-Omicron Subpopulations.
  * For participants without variant information, those randomized under Protocol v7 on or after December 15, 2021 would be assigned to the Omicron Subpopulation, and those randomized on or before December 14, 2021 would be assigned to the Non-Omicron Subpopulation.
  CASIRIVIMAB + IMDEVIMAB: 600 mg casirivimab and 600 mg imdevimab, administered together as single IV infusion as one-time dose at study entry. Participants are no longer being randomized to this intervention.
- Camostat (Phase 2): Administered as oral tablets Camostat: 200 mg (2 x 100 mg) film-coated tablets administered orally every 6 hours for 7 days. Participants are no longer being randomized to this intervention.
- SNG001 (Phase 2): Administered by inhalation SNG001: 1.3 mL solution administered once daily for 14 days using Aerogen Ultra nebulizer (inhalation device). Participants are no longer being randomized to this intervention.
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 383 | 397 | 55 | 51 | 103 | 111 | 0 | 0 | 121 | 134 | 0 | 0 | 105 | 107 | 198 | 194 | 0 | 0 | 0 | 0
Days |  |  |  |  |  | 19.0 [16.0 to 23.0] | 23.0 [19.0 to 25.0] | 16.00 [11.00 to 22.00] | 17.00 [11.00 to 23.00] | 16.00 [14.00 to 18.00] | 14.00 [12.00 to 17.00] |  |  | 16.0 [15.0 to 21.0] | 24.0 [17.0 to NA] — The upper confidence interval from the Kaplan-Meier product-limit-estimates is not available as there are not enough events during the later timepoints in the study. Consequently, the median and/or confidence limit could not be statistically estimated. |  |  | 8.0 [6.0 to 10.0] | 10.0 [8.0 to 13.0] | 18.0 [16.0 to 21.0] | NA [20.0 to NA] — The median and upper confidence interval from the Kaplan-Meier product-limit-estimates are not available as there are not enough events beyond the halfway timepoint in the study. Consequently, the median and/or confidence limit could not be statistically estimated. |  |  |  |

15. Secondary Outcome: COVID-19 Symptom Severity Ranking (Phases 2 and 3)
Description: Symptoms scored daily as absent (score 0), mild (score 1), moderate (score 2) or severe (score 3). Symptoms: feeling feverish, cough, shortness of breath/difficulty breathing at rest/with activity, sore throat, body pain/muscle pain/aches, fatigue, headache, chills, nasal obstruction/congestion, nasal discharge, nausea, vomiting, and diarrhea. Subjects alive and never hospitalized through Day 28: Symptom Severity Ranking=subject-specific AUC (area under curve) joining daily total symptom score associated with COVID-19 disease, over time (through Day 28, counting Day 0 as first day), calculated by trapezoidal rule and rescaled for time by dividing by the total number of trapezoids. Subjects who died within Day 28: Assigned severity score 42; Subjects alive but remaining hospitalized at Day 28: Assigned severity score 41; Subjects alive but no longer hospitalized at Day 28: Assigned severity score 40.
  Calculated Severity Score=scale of 0 to 42. Higher value=worse health condition.
Time Frame: From Day 0 thru Day 28
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Mean (Standard Deviation); unit: units on a scale*days
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Placebo (Phase 2)
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 990 | 383 | 397 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 198 | 194 | 121 | 134 | 107 | 102 | 105 | 107
units on a scale*days | 3.4940 (7.83544) | 5.6939 (11.09572) | 4.1395 (7.35047) | 4.0378 (7.37122) | 4.4001 (7.42311) | 4.1213 (6.12801) | 7.8505 (12.16647) | 3.5 (3.35) | 5.8 (10.44) | 4.6 (8.16) | 5.5 (9.74) | 3.6360 (4.67064) | 5.5345 (9.68874) | 5.3314 (9.41155) | 5.1306 (8.69588) | 4.1020 (6.33252) | 4.5759 (7.82761) | 4.7658 (6.71588) | 5.0532 (6.03326) | 5.6263 (8.89389) | 4.5862 (6.27948) | 4.6631 (8.38511) | 4.5728 (7.87041) | 4.6 (7.51) | 4.2 (6.88)

16. Secondary Outcome: Proportion of Participants With ≥1 Worsening Symptom of COVID-19 (Phases 2 and 3)
Description: Progression of one or more COVID-19-associated symptoms to a worse status than recorded in study diary at study entry, prior to start of investigational product or placebo
Time Frame: Thru Day 28
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 990 | 383 | 397 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Participants | 42 | 40 | 102 | 105 | 876 | 323 | 321 | 42 | 43 | 87 | 96 | 86 | 92 | 82 | 92 | 81 | 81 | 102 | 119 | 83 | 79 | 70 | 86 | 160 | 157

17. Secondary Outcome: Time to Self-reported Return to Usual Health (a) (Phases 2 and 3)
Description: Defined as the number of days from start of investigational treatment until the first of two consecutive days that a participant reported return to usual (pre-COVID-19) health as recorded in a participant's study diary.
  Not analyzed for Bamlanivimab Phase 2 and Phase 3 arms.
Time Frame: Thru Day 28
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  This OM was not a pre-specified outcome for all Bamlanivimab arms (Phase 2 & 3) and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Bamlanivimab 7000mg Placebo (Phase 2): Administered by IV infusion Placebo for Bamlanivimab 7000mg: Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
- Bamlanivimab 700mg (Phase 2); Bamlanivimab 700mg (Phase 3): Administered by IV infusion bamlanivimab 700mg: Administered by single IV infusion. Participants are no longer being randomized to this intervention.
- Bamlanivimab 700mg Placebo (Phase 2): Administered by IV infusion Placebo for Bamlanivimab 700mg: Commercially available 0.9% sodium chloride solution. Participants are no longer being randomized to this intervention.
Arm/Group | Bamlanivimab 7000mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 383 | 397 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Days |  |  |  |  |  | 16.0 [14.0 to 19.0] | 22.0 [18.0 to 26.0] | 11.00 [7.00 to 15.00] | 15.00 [8.00 to 19.00] | 14.00 [8.00 to 16.00] | 13.00 [11.00 to 16.00] | 19.0 [17.0 to 24.0] | 17.0 [13.0 to 19.0] | 12.0 [10.0 to 16.0] | 14.0 [11.0 to 17.0] | 15.0 [12.0 to 21.0] | 17.0 [14.0 to 22.0] | 11.0 [10.0 to 15.0] | 12.0 [9.0 to 17.0] | 12.0 [9.0 to 18.0] | 17.0 [14.0 to 21.0] | 12.0 [10.0 to 16.0] | 17.0 [12.0 to 19.0] | 15.0 [12.0 to 18.0] | 13.0 [10.0 to 16.0]

18. Secondary Outcome: Cumulative Incidence of Death Due to Any Cause or Hospitalization Due to Any Cause (Phases 2 and 3)
Description: as for outcome 6
Time Frame: Day 0 thru Week 24
Population: as for outcome 15
Measure: Number; unit: Events
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 990 | 383 | 397 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Events | 2 | 4 | 5 | 5 | 44 | 13 | 46 | 1 | 5 | 5 | 8 | 2 | 7 | 6 | 6 | 3 | 5 | 7 | 8 | 5 | 5 | 7 | 5 | 6 | 5

19. Secondary Outcome: Cumulative Incidence of Death Due to Any Cause or Hospitalization Due to Any Cause (Phases 2 and 3)
Description: Not applicable to Bamlanivimab arms as these were only 24 week-long studies. Hospitalization defined as ≥24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address medical needs of those with severe COVID-19. An event is defined as first occurrence of hospitalization/death (i.e. if subject has multiple hospitalizations, only the first hospitalization is counted as an event). Therefore, an event can only occur once for a subject. Results are presented as number of events.
Time Frame: Day 0 thru Week 72
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  All Bamlanivimab arms (Phase 2 & 3) were only 24 week-long studies, therefore this OM was not a pre-specified outcome and is not applicable.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Number; unit: Events
Groups:
- Bamlanivimab 7000 mg (Phase 2): Administered by IV infusion. bamlanivimab 7000mg: Administered by single IV infusion. Participants are no longer being randomized to this intervention.
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 383 | 397 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Events |  |  |  |  |  | 23 | 59 | 3 | 5 | 7 | 8 | 2 | 7 | 9 | 6 | 4 | 5 | 11 | 9 | 5 | 5 | 7 | 5 | 10 | 13

20. Secondary Outcome: Oxygen Saturation Level (Phases 2 and 3)
Description: Measured by pulse oximeter and categorized as <96% versus ≥96%. Analysis not performed for Bamlanivimab arms.
Time Frame: Thru Day 28
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 106 | 101 | 45 | 44 | 91 | 93 | 100 | 97 | 90 | 91 | 98 | 92 | 106 | 119 | 98 | 91 | 89 | 90 | 182 | 178
Participants
  Oxygen Saturation ≥96% |  |  |  |  |  | 94 | 94 | 45 | 42 | 89 | 90 | 99 | 95 | 87 | 87 | 95 | 90 | 97 | 111 | 96 | 89 | 88 | 88 | 177 | 171
  Oxygen Saturation <96% |  |  |  |  |  | 12 | 7 | 0 | 2 | 2 | 3 | 1 | 2 | 3 | 4 | 3 | 2 | 9 | 8 | 2 | 2 | 1 | 2 | 5 | 7
  Missing pulse oximetry records: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 10 | 7 | 12 | 18 | 10 | 13 | 16 | 13 | 98 | 92 | 106 | 119 | 98 | 91 | 89 | 90 | 182 | 178
  Missing pulse oximetry records |  |  |  |  |  | 6 | 7 | 10 | 7 | 12 | 18 | 10 | 13 | 16 | 13 | 6 | 11 | 15 | 15 | 9 | 11 | 16 | 17 | 16 | 13

21. Secondary Outcome: AUC of SARS-CoV-2 RNA From Site-collected NP Swabs (Phase 2)
Description: Measured by area under the curve (AUC) and above assay lower limit of quantification of quantitative SARS-CoV-2 RNA over time.
  Not analyzed for Bamlanivimab arms.
Time Frame: Thru Day 14
Population: Analysis population description (Phase 2): mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Participants with missing or unsuitable samples were excluded from analysis. All placebo arms except for Bamlanivimab include pooled placebo data. This OM was not a pre-specified outcome for Bamlanivimab Phase 2 and therefore not done.
Measure: Mean (Standard Deviation); unit: units on a scale*days
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 46 | 87 | 95 | 105 | 100 | 96 | 84 | 96 | 96 | 99 | 94 | 100 | 100
units on a scale*days |  |  |  |  | 9.2 (10.127) | 11.7 (16.505) | 12.5 (11.497) | 14.0 (15.134) | 13.7450 (11.03930) | 13.1472 (13.34285) | 15.2756 (12.81071) | 13.9833 (13.85182) | 11.2405 (12.06870) | 12.8663 (14.03668) | 11.6766 (11.40875) | 13.6064 (14.17869) | 9.5 (11.20) | 10.9 (11.87)

22. Secondary Outcome: Proportion of Participants With New Adverse Event (AE) ≥ Grade 2 (Phases 2 and 3)
Time Frame: Thru Day 28
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Bamlanivimab Phase 3 enrolled under Protocol v1, this OM was a new addition in v7 for Phase 3 so this OM was not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 0 | 112 | 109 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Participants | 19 | 16 | 47 | 30 |  | 29 | 45 | 20 | 14 | 30 | 25 | 24 | 31 | 29 | 25 | 20 | 26 | 40 | 45 | 25 | 23 | 22 | 28 | 58 | 60

23. Secondary Outcome: Proportion of Participants With New Adverse Event (AE) ≥ Grade 2 (Phases 2 and 3)
Time Frame: Thru Week 24
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Bamlanivimab 700mg (Phase 3) enrolled under Protocol v1, this OM was a new addition in v7 for Phase 3 so this OM was not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 48 | 46 | 111 | 112 | 0 | 112 | 109 | 55 | 51 | 103 | 111 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 105 | 107 | 198 | 194
Participants | 22 | 18 | 53 | 39 |  | 45 | 50 | 23 | 17 | 38 | 33 | 34 | 41 | 32 | 32 | 27 | 32 | 46 | 60 | 31 | 30 | 76 | 74 | 72 | 69

24. Secondary Outcome: Proportion of Participants With New Adverse Event (AE) ≥ Grade 3 (Phases 2 and 3)
Time Frame: Thru Week 24
Population: Analysis population description: mITT analysis set = randomized and treated = all with randomization date - (randomized not treated + screen fail but randomized + excluded from analyses at NIH request + dual enrolled subject).
  Bamlanivimab Ph2 enrolled under Protocol v1, AZD7442, BMS enrolled under v6, this OM was a new addition for Phase 2 agents in v7 so this OM was not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Count of Participants; unit: Participants
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 990 | 383 | 397 | 0 | 0 | 0 | 0 | 110 | 110 | 106 | 105 | 106 | 103 | 121 | 134 | 107 | 102 | 0 | 0 | 198 | 194
Participants |  |  |  |  | 92 | 37 | 74 |  |  |  |  | 5 | 11 | 12 | 12 | 8 | 13 | 17 | 27 | 11 | 12 |  |  | 30 | 18

25. Secondary Outcome: Time to Self-reported Return to Usual Health (b) (Phases 2 and 3)
Description: Defined as the number of days from start of investigational treatment until the first of four consecutive days that a participant reported return to usual (pre-COVID-19) health as recorded in a participant's study diary.
  Not collected for Bamlanivimab Phase 2 and Phase 3 arms.
Time Frame: Thru Day 28
Population: Analysis population description: Number of subjects in analysis = participants who returned to usual (pre-COVID-19) health.
  Bamlanivimab Phase 2&3 enrolled under v1, Camostat, SNG001, BRII, SAB Ph2 enrolled under Protocol v6 or earlier, OM was new addition in Protocol v8, not pre-specified and therefore not done.
  BRII-196+BRII-198 Placebo includes pooled placebo data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 55 | 51 | 103 | 111 | 0 | 0 | 121 | 134 | 0 | 0 | 105 | 107 | 198 | 194 | 0 | 0 | 0 | 0
Days |  |  |  |  |  |  |  | 13.00 [9.00 to 21.00] | 17.00 [9.00 to 21.00] | 15.00 [11.00 to 19.00] | 15.00 [12.00 to 18.00] |  |  | 14.0 [10.0 to 16.0] | 15.0 [10.0 to 19.0] |  |  | 13.0 [10.0 to 17.0] | 17.0 [13.0 to 23.0] | 17.0 [15.0 to 20.0] | 15.0 [12.0 to 18.0] |  |  |  |

ADVERSE EVENTS:
Time Frame: Week 24 for Bamlanivimab arms. Week 72 for all other arms.
Description: Safety Analysis Set: randomized and treated=all with randomization date - (randomized not treated+screen fail but randomized+excluded from analyses at NIH request+dual enrolled subject). Summarized by actual treatment received.
  8 participants allocated to BRII Placebo arm received active treatment. Pooled placebo except Bamlanivimab, SAB (Phase 3) and Casirivimab+Imdevimab (Phase 3) arms.
  SAEs=Serious Treatment Emergent Adverse Events (TEAEs) Other (non-Serious) AEs=Other (non-Serious) TEAEs
Arm/Group | Bamlanivimab 7000 mg (Phase 2) | Bamlanivimab 7000mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 2) | Bamlanivimab 700mg Placebo (Phase 2) | Bamlanivimab 700mg (Phase 3) | BRII-196+BRII-198 (Pooled Phase 2/3) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) | AZD7442 (IV) (Phase 2) | AZD7442 (IV) Pooled Placebo (Phase 2) | AZD7442 (IM) (Phase 2) | AZD7442 (IM) Pooled Placebo (Phase 2) | SNG001 (Phase 2) | SNG001 Pooled Placebo (Phase 2) | Camostat (Phase 2) | Camostat Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 2) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) | SAB-185 (Low Dose) (Phase 3) OMICRON Population | Casirivimab and Imdevimab (Phase 3) OMICRON Population | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population | SAB-185 (High Dose) (Phase 2) | SAB-185 (High Dose) Pooled Placebo (Phase 2) | BMS 986414+BMS 986413 (Phase 2) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/46 | 0/111 | 0/112 | 12/990 | 2/383 | 11/397 | 0/55 | 1/51 | 0/103 | 1/111 | 0/110 | 0/110 | 1/106 | 1/105 | 0/106 | 0/103 | 1/198 | 4/194 | 4/121 | 1/134 | 0/107 | 0/102 | 0/105 | 0/107
Serious Adverse Events (participants affected / at risk) | 2/48 | 6/46 | 5/111 | 4/112 | 57/990 | 25/390 | 56/390 | 0/55 | 4/51 | 4/103 | 7/111 | 2/110 | 8/110 | 9/106 | 7/105 | 5/106 | 5/103 | 10/198 | 13/194 | 11/121 | 10/134 | 5/107 | 5/102 | 7/105 | 5/107
Other Adverse Events (participants affected / at risk) | 26/48 | 26/46 | 69/111 | 57/112 | 334/990 | 223/390 | 228/390 | 29/55 | 20/51 | 40/103 | 40/111 | 54/110 | 57/110 | 53/106 | 57/105 | 52/106 | 42/103 | 93/198 | 91/194 | 64/121 | 85/134 | 59/107 | 40/102 | 52/105 | 48/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bamlanivimab 7000 mg (Phase 2) (N=48) | Bamlanivimab 7000mg Placebo (Phase 2) (N=46) | Bamlanivimab 700mg (Phase 2) (N=111) | Bamlanivimab 700mg Placebo (Phase 2) (N=112) | Bamlanivimab 700mg (Phase 3) (N=990) | BRII-196+BRII-198 (Pooled Phase 2/3) (N=390) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) (N=390) | AZD7442 (IV) (Phase 2) (N=55) | AZD7442 (IV) Pooled Placebo (Phase 2) (N=51) | AZD7442 (IM) (Phase 2) (N=103) | AZD7442 (IM) Pooled Placebo (Phase 2) (N=111) | SNG001 (Phase 2) (N=110) | SNG001 Pooled Placebo (Phase 2) (N=110) | Camostat (Phase 2) (N=106) | Camostat Pooled Placebo (Phase 2) (N=105) | SAB-185 (Low Dose) (Phase 2) (N=106) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) (N=103) | SAB-185 (Low Dose) (Phase 3) OMICRON Population (N=198) | Casirivimab and Imdevimab (Phase 3) OMICRON Population (N=194) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population (N=121) | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population (N=134) | SAB-185 (High Dose) (Phase 2) (N=107) | SAB-185 (High Dose) Pooled Placebo (Phase 2) (N=102) | BMS 986414+BMS 986413 (Phase 2) (N=105) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 17 | 6 | 38 | 0 | 3 | 4 | 6 | 1 | 7 | 4 | 4 | 1 | 4 | 3 | 3 | 6 | 2 | 1 | 4 | 3 | 4
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serratia bacteremia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug use disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder perforation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture blisters (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Physical assault (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bamlanivimab 7000 mg (Phase 2) (N=48) | Bamlanivimab 7000mg Placebo (Phase 2) (N=46) | Bamlanivimab 700mg (Phase 2) (N=111) | Bamlanivimab 700mg Placebo (Phase 2) (N=112) | Bamlanivimab 700mg (Phase 3) (N=990) | BRII-196+BRII-198 (Pooled Phase 2/3) (N=390) | BRII-196+BRII-198 Placebo (Pooled Phase 2/3) (N=390) | AZD7442 (IV) (Phase 2) (N=55) | AZD7442 (IV) Pooled Placebo (Phase 2) (N=51) | AZD7442 (IM) (Phase 2) (N=103) | AZD7442 (IM) Pooled Placebo (Phase 2) (N=111) | SNG001 (Phase 2) (N=110) | SNG001 Pooled Placebo (Phase 2) (N=110) | Camostat (Phase 2) (N=106) | Camostat Pooled Placebo (Phase 2) (N=105) | SAB-185 (Low Dose) (Phase 2) (N=106) | SAB-185 (Low Dose) Pooled Placebo (Phase 2) (N=103) | SAB-185 (Low Dose) (Phase 3) OMICRON Population (N=198) | Casirivimab and Imdevimab (Phase 3) OMICRON Population (N=194) | SAB-185 (Low Dose) (Phase 3) Non-OMICRON Population (N=121) | Casirivimab and Imdevimab (Phase 3) Non-OMICRON Population (N=134) | SAB-185 (High Dose) (Phase 2) (N=107) | SAB-185 (High Dose) Pooled Placebo (Phase 2) (N=102) | BMS 986414+BMS 986413 (Phase 2) (N=105) | BMS 986414+BMS 986413 Pooled Placebo (Phase 2) (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Granulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoconcentration (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nucleated red cells (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atroventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left atrial enlargement (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 3 | 0 | 3 | 4 | 8 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 1 | 0 | 4 | 0 | 3 | 0 | 2 | 1 | 4 | 0 | 5
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermobility syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tourette's disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastoid disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Graves' disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Holmes-Adie pupil (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 5 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 3 | 6 | 25 | 21 | 14 | 3 | 0 | 5 | 4 | 13 | 6 | 8 | 5 | 6 | 1 | 6 | 5 | 4 | 6 | 6 | 1 | 5 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 5 | 6 | 17 | 10 | 13 | 3 | 2 | 2 | 3 | 6 | 4 | 8 | 5 | 1 | 4 | 4 | 5 | 4 | 8 | 4 | 4 | 3 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 2 | 9 | 5 | 1 | 2 | 0 | 1 | 2 | 1 | 3 | 2 | 2 | 2 | 3 | 2 | 3 | 4 | 2 | 2 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Application site hyperaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 2 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Chills (General disorders) | 1 | 1 | 4 | 4 | 8 | 7 | 8 | 0 | 0 | 2 | 2 | 7 | 4 | 1 | 2 | 0 | 1 | 7 | 4 | 4 | 6 | 2 | 1 | 2 | 2
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehiscence (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 8 | 2 | 16 | 16 | 22 | 2 | 3 | 2 | 3 | 11 | 6 | 7 | 7 | 3 | 2 | 13 | 9 | 8 | 9 | 8 | 2 | 7 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site paraesthesia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion stie pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1 | 4 | 5 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 6 | 1 | 6 | 6 | 8 | 0 | 1 | 1 | 2 | 8 | 4 | 9 | 1 | 4 | 2 | 4 | 5 | 4 | 6 | 5 | 2 | 2 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Physical deconditioning (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 8 | 1 | 19 | 11 | 8 | 1 | 2 | 0 | 2 | 6 | 3 | 3 | 3 | 1 | 1 | 7 | 7 | 7 | 6 | 2 | 1 | 3 | 1
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunodeficiency common variable (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iodine allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 7 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 0 | 2 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicitis gonococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 33 | 25 | 0 | 0 | 0 | 0 | 21 | 10 | 12 | 14 | 13 | 4 | 8 | 7 | 9 | 15 | 6 | 4 | 10 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 3 | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Monkeypox (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mycobacterium kansasii infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 13 | 11 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 1 | 1 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Root canal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 7 | 5 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 3 | 4 | 2 | 4 | 0 | 1 | 0 | 2
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 5 | 10 | 9 | 2 | 0 | 0 | 1 | 5 | 2 | 3 | 3 | 4 | 1 | 2 | 3 | 1 | 5 | 1 | 1 | 5 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 8 | 9 | 6 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 3 | 1 | 3 | 0 | 2 | 2 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 2 | 13 | 5 | 4 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 2 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3 | 4 | 9 | 4 | 14 | 3 | 2 | 5 | 3 | 4 | 10 | 8 | 2 | 5 | 9 | 5 | 3 | 4 | 3 | 2 | 8 | 4 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 4 | 3 | 8 | 1 | 2 | 1 | 2 | 2 | 7 | 3 | 2 | 1 | 6 | 2 | 2 | 2 | 3 | 0 | 5 | 3 | 6
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biopsy cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood acid phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 3 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
Blood bilirubin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 4 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1
Blood bilirubin unconjugated decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2
Blood creatinine increased (Investigations) | 2 | 2 | 1 | 1 | 2 | 7 | 6 | 1 | 3 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 15 | 12 | 3 | 2 | 4 | 0 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 3 | 0 | 4 | 4 | 35 | 18 | 18 | 4 | 2 | 9 | 4 | 1 | 8 | 4 | 4 | 6 | 3 | 21 | 20 | 10 | 15 | 5 | 2 | 6 | 5
Blood iron decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood osmolarity increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 4 | 2 | 2 | 5 | 6 | 6 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Blood sodium abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 6 | 3 | 2 | 1 | 1 | 0 | 4 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea nitrogen/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood zinc decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature fluctuation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coagulation test abnormal (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 11 | 0 | 1 | 2 | 0 | 1 | 4 | 2 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 3 | 1 | 2
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Differential white blood cell count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 10 | 0 | 0 | 3 | 0 | 0 | 4 | 2 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 1
Full blood count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Globulins increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 2 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Grip strength decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Haematocrit increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 2 | 3 | 2 | 2 | 7 | 0 | 1 | 1 | 1 | 3 | 5 | 2 | 2 | 0 | 4 | 1 | 3 | 3 | 0 | 1 | 4 | 0 | 2
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
High density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HIV test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immature granulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 2 | 0 | 1 | 4 | 2 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 3 | 1 | 2
Red cell distribution width increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 8 | 0 | 1 | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Transferrin saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 2 | 6 | 5 | 0 | 0 | 0 | 1 | 4 | 5 | 0 | 3 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 6 | 9 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 4 | 5 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 13 | 6 | 14 | 0 | 2 | 2 | 2 | 0 | 2 | 2 | 1 | 3 | 6 | 5 | 4 | 1 | 2 | 3 | 5 | 2 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 1 | 2 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0 | 7 | 15 | 17 | 0 | 2 | 0 | 3 | 4 | 8 | 2 | 9 | 2 | 3 | 3 | 5 | 1 | 5 | 3 | 2 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 8 | 7 | 9 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 5 | 3 | 1 | 0 | 3 | 4 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 9 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 1 | 2 | 1 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5 | 1 | 6 | 4 | 9 | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 2 | 3 | 1 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 8 | 4 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 2 | 2 | 6 | 6 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 7 | 9 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 2 | 5 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 1 | 1
Anosmia (Nervous system disorders) | 0 | 2 | 3 | 3 | 9 | 7 | 4 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 2 | 1 | 3 | 7 | 6 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 1 | 2 | 2 | 2 | 0 | 0 | 3 | 4 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 3 | 8 | 8 | 9 | 1 | 0 | 1 | 2 | 5 | 4 | 2 | 4 | 1 | 2 | 1 | 3 | 0 | 5 | 6 | 1 | 2 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 6 | 8 | 9 | 29 | 31 | 34 | 4 | 2 | 4 | 2 | 11 | 10 | 9 | 6 | 2 | 7 | 3 | 5 | 4 | 8 | 6 | 7 | 4 | 5
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Morton's neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 2 | 1 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulnar nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Labour pain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abulia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 3 | 5 | 5 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 3 | 1 | 3 | 0 | 1 | 1 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Borderline personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired reasoning (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 1 | 5 | 16 | 12 | 1 | 1 | 1 | 3 | 4 | 3 | 3 | 3 | 1 | 0 | 0 | 2 | 2 | 2 | 7 | 0 | 3 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Terminal insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tobacco abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 0 | 1 | 0 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile dermatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 0 | 17 | 17 | 17 | 1 | 1 | 6 | 3 | 12 | 7 | 7 | 6 | 3 | 2 | 7 | 8 | 8 | 11 | 3 | 2 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6 | 8 | 14 | 7 | 19 | 1 | 0 | 7 | 2 | 11 | 7 | 6 | 4 | 3 | 2 | 7 | 6 | 11 | 12 | 3 | 2 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 6 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 4 | 7 | 7 | 7 | 1 | 0 | 1 | 0 | 4 | 3 | 3 | 3 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 4 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 9 | 3 | 4 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 7 | 5 | 6 | 5 | 2 | 1 | 2 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal cobble stone mucosa (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 3 | 9 | 10 | 16 | 1 | 0 | 3 | 0 | 6 | 4 | 5 | 2 | 4 | 4 | 4 | 3 | 3 | 4 | 6 | 4 | 4 | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 12 | 8 | 6 | 2 | 0 | 3 | 1 | 4 | 6 | 5 | 4 | 1 | 1 | 7 | 4 | 4 | 6 | 4 | 1 | 3 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 7 | 10 | 10 | 1 | 0 | 0 | 0 | 3 | 8 | 2 | 4 | 3 | 3 | 1 | 2 | 2 | 5 | 8 | 3 | 3 | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture blisters (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 4 | 2 | 5 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 2 | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria cholinergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Victim of crime (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial insufficiency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 4 | 4 | 11 | 15 | 18 | 1 | 1 | 3 | 2 | 3 | 4 | 4 | 5 | 5 | 3 | 8 | 9 | 7 | 13 | 5 | 3 | 2 | 5
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (8):
  • Study Protocol and Informed Consent Form: Protocol v8.0 (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/Prot_ICF_004.pdf
  • Study Protocol and Informed Consent Form: Letter of Amendment 1 for Protocol v8.0 (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/Prot_ICF_005.pdf
  • Statistical Analysis Plan: Primary SAPs v1.0-v10.0 (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/SAP_006.pdf
  • Statistical Analysis Plan: SAPs for Phase 2 and 3 CSRs v1.0-v5.0 (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/SAP_007.pdf
  • Informed Consent Form: Multiple Study Drugs Site ICF 1 (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/ICF_001.pdf
  • Informed Consent Form: Optional Extra Samples ICF (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/ICF_002.pdf
  • Informed Consent Form: Study Drug LY3819253 (Bamlanivimab) ICF (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/ICF_003.pdf
  • Informed Consent Form: Multiple Study Drugs Site ICF 2 (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04518410/ICF_008.pdf